

| Study | <b>Protocol</b> |
|-------|-----------------|
| Stuay | Protocor |

Study Code D2287R00166

Version 7.4

Date August 10, 2021

# Managing Asthma Patients with AMAZE<sup>TM</sup>: A Novel Disease Management Platform, A Clinical Pilot Study

Sponsor:
AstraZeneca Pharmaceuticals, LP

PPD
PPD
PPD

#### TABLE OF CONTENTS 2 TITLE PAGE ....... 1 TABLE OF CONTENTS......2 RESPONSIBLE PARTIES......7 AMENDMENT HISTORY ......13 1. BACKGROUND AND RATIONALE......15 1.1 1.2 OBJECTIVES AND HYPOTHESES......15 2. 2.1 2.2 Secondary Objective(s) and Hypothesis(es) (Optional)......16 2.3 METHODOLOGY ......16 3. 3.1 3.1.1 3.2 3.3 3.4 Exclusion Criteria 19 VARIABLES AND EPIDEMIOLOGICAL MEASUREMENTS ......19 4. 4.1 Patient-Completed......21 4.1.1 AMAZE<sup>TM</sup> Patient App ......21 4.1.1.1 4.1.1.2 4.1.1.3 4.1.1.4 Patient Visit Experience Survey ......21 4.1.1.5 System Usability Scale ......22 4.1.1.6 PSO-18......22 4.1.1.7 4.1.2

Study Protocol Form Version 7.4

4.1.2.1

Form Doc ID: AZDoc0059948

Parent Doc ID: SOP LDMS\_001\_001643282

| 4.1.2.2 | Chart Review Case Report Form | .23 |
|---|---|---|
| 4.1.2.3 | System Usability Scale | |
| 4.1.2.4 | Post-study Survey | .23 |
| 4.2 | Outcomes | 23 |
| 4.2.1 | Primary Outcome | |
| 4.2.2 | Secondary Outcome | |
| 4.2.3 | Exploratory Outcome One | |
| 4.2.4 | Exploratory Outcome Two | |
| 4.3 | Other Variables and Covariates | |
| 5. | STATISTICAL ANALYSIS PLAN | .25 |
| 5.1 | Statistical Methods: General Aspects | 25 |
| 5.1.1 | Primary Objective: To generate evidence on the feasibility, usability, | .23 |
| 3.1.1 | perceived value, and potential benefits of the AMAZE <sup>TM</sup> implemented in | |
| | clinical practice | 25 |
| 5.1.2 | Secondary Objective(s) | |
| 5.1.3 | Exploratory Objective One: To assess how the implementation of AMAZE <sup>TM</sup> | .23 |
| 5.1.5 | affects clinical outcomes | 25 |
| 5.1.4 | Exploratory Objective Two: To identify patients who are most likely to benefit | |
| 0.11. | from using AMAZE <sup>TM</sup> | |
| <i>5</i> 2 | | |
| 5.2 | Bias | |
| 5.2.1 | Methods to Minimize Bias | |
| 5.2.2<br>5.2.3 | Adjustment for Multiple Comparisons | |
| | Strengths and Limitations | |
| 5.3 | Sample Size and Power Calculations | |
| 6. | STUDY CONDUCT AND REGULATORY DETAILS | .26 |
| 6.1 | Study Conduct | .26 |
| 6.1.1 | Procedures | .26 |
| 6.1.1.1 | Recruitment | |
| 6.1.1.2 | Baseline Visit | |
| 6.1.1.3 | Longitudinal Follow-up Interviews and Assessments | |
| 6.1.1.4 | Cross-Sectional Follow-up Interviews and Assessments | |
| 6.1.1.5 | Claims Data Export | |
| 6.1.2 | Quality Control | |
| 6.1.2.1 | Monitoring | |
| 6.1.2.2 | Contacts with the sites to: | |
| 6.1.2.3 | Remote Monitoring activities for: | |
| 6.1.2.4 | Training of Study Site Personnel | |
| 6.1.2.5 | ePRO Programming and Hosting | |
| 6.2 | Protection of Human Subjects | .30 |
| 6.2.1 | Informed Consent | |
| 6.2.2 | Confidentiality of Study/Patient Data | .31 |

| 6.3 | Collection and Reporting of Adverse Events/Adverse Drug Reactions | 32 |
|---|---|---|
| 6.3.1 | Collection of Adverse Events | |
| 6.3.2<br>6.3.3 | Reporting of Adverse Events | |
| 7. | Aggregate Safety Review from PRO Instruments | |
| 8. | APPENDIX A. PATIENT SCREENING SCRIPT | |
| 9. | APPENDIX B. ELECTRONIC CONSENT EMAIL | |
| 10. | APPENDIX C. RECRUITMENT EMAIL AND FLYER | |
| 11. | APPENDIX D. INTRODUCTORY EMAIL | 43 |
| 12. | APPENDIX E. AMAZE <sup>TM</sup> PATIENT MOBILE APPLICATION SCREENSHOTS | 44 |
| 12.1 | Flyer for App | 44 |
| 12.2 | Account Creation and Login | 45 |
| 12.3 | Terms of Use | 49 |
| 12.4 | Air Quality | 51 |
| 12.5 | Appointments | 53 |
| 12.6 | Asthma Control Test | 54 |
| 12.7 | Daily Asthma Log | 59 |
| 12.8 | Education | |
| 12.9 | Email Password Reset | 67 |
| 12.10 | Home | 68 |
| 12.11 | Messages | 69 |
| 12.12 | Feedback | |
| 12.13 | My Plan | 73 |
| 12.14 | Notifications | 76 |
| 12.15 | Settings | 77 |
| 12.16 | Trends | 81 |
| 12.17 | Study Ending | 85 |
| 13. | APPENDIX F. CLINICAL CASE REPORT FORM | 87 |
| 14. | APPENDIX G. PATIENT DEMOGRAPHIC QUESTIONNAIRE | 91 |
| 15. | APPENDIX H. PATIENT VISIT EXPERIENCE SURVEY | 95 |
| 16. | APPENDIX I. POST-STUDY SURVEY (FOR HCPS) | |
| 17.<br>Study Proto | APPENDIX J. PATIENT SATISFACTION QUESTIONNAIRE-18 (PSQ | |

| 18. | APPENDIX K. SIX-MONTH CHART REVIEW CASE REPORT FORM | 104 |
|---|---|---|
| 20. | APPENDIX L. MGH WORKFLOW FOR IMPLEMENTATION OF DMP IN CLINICAL PRACTICE. | |
| 21. | APPENDIX M. PATIENT USER EXPERIENCE SURVEY | 110 |
| 22. | APPENDIX N.1 SYSTEM USABILITY SCALE (SUS) ADMINISTERED AT MONTHS 1 AND 6: Patients | 114 |
| 23. | APPENDIX N.2 SYSTEM USABILITY SCALE (SUS) ADMINISTERED AT MONTHS 1 AND 6: MGH Staff | 115 |
| 24. | APPENDIX O. FOLLOW-UP SEMI-STRUCTURED INTERVIEW GUIDES | 116 |
| 25. | APPENDIX P. RECRUITMENT TRACKING LOG | 124 |
| 26. | SIGNATURES | 126 |

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| Abbreviation or special term | Explanation |
|---|---|
| ACTTM | Asthma Control Test |
| AE | Adverse event |
| AZ | AstraZeneca |
| CFR | Code of Federal Regulations |
| COPD | Chronic obstructive pulmonary disease |
| CRF | Case report form |
| CRO | Clinical research organization |
| DES | Data entry site |
| EMR | Electronic medical record |
| ePRO | Electronic patient-reported outcome |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HCP | Healthcare practitioner |
| HIPAA | Health Insurance Portability and Accountability Act |
| ICH | International Council for Harmonization |
| ICS | Inhaled corticosteroid |
| ID | Identifier |
| IEC | Independent Ethics Committee |
| IRB | Institutional review board |
| LABA | Long-acting beta agonist |
| MC | Marketing company |
| MEOR | Medical Evidence and Observational Research |
| MGH | Massachusetts General Hospital |
| OCR | Optical character recognition |
| SD | Standard deviation |
| SOP | Standard operating procedure |
| SUA | Severe uncontrolled asthma |

# **RESPONSIBLE PARTIES**

| Name | Professional Title | Role in<br>Study | Affiliation | Email Address |
|---|---|---|---|---|
| PPD | PPD US Respiratory Medical | Team Lead | AstraZeneca | PPD |
| PPD | PPD | Medical Lead | AstraZeneca | PPD |
| PPD | PPD Patient-Centered Research | Senior Advisor | Evidera | PPD |
| Elizabeth<br>Bacci | Research Scientist | Principal<br>Investigator | Evidera | PPD |
| PPD | PPD | Site<br>Investigator | MGH | PPD |
| PPD | Pulmonary and Critical<br>Care Medicine | Site<br>Investigator | MGH | PPD |
| PPD | PPD Pediatric Pulmonary Unit | Site<br>Investigator | MGH | PPD |
| PPD | PPD Health<br>Information<br>Technology | Production<br>Team Lead | AstraZeneca | PPD |

#### PROTOCOL SYNOPSIS

AMAZE<sup>TM</sup> Asthma Implementation Clinical Pilot Study: MGH

Background/Rationale: AstraZeneca (AZ) has developed the AMAZE<sup>TM</sup> disease management platform to be used across multiple disease indications to provide a unified experience for the management of patients throughout their patient care journey. AMAZE<sup>TM</sup> integrates multiple systems, including a patient Application where patients can enter daily symptoms and impact to communicate this information to their healthcare provider (HCP), as well as access disease educational materials. Both the patient Application and a clinician dashboard are integrated with the patient's electronic medical records (EMR) to provide a clear view of the patient's health status both in and out of the clinic. Implementation of AMAZE<sup>TM</sup> within clinical practice has not yet been evaluated. The results from this study will be used to inform any changes or modifications that need to be made to the technology platform, its implementation process, and explore impact on clinical outcomes.

#### **Objectives and Hypotheses:**

The primary study objective is to generate evidence as to the feasibility, usability, perceived value, and potential benefits of implementing the AMAZE<sup>TM</sup> platform into clinical practice. This objective will be accomplished through the generation of evidence in two key outcome types:

- 1. **Technology Outcomes**: Key questions to be asked regarding the technology outcomes are:
  - How much is the platform utilized, and what is the perceived value by both clinical staff and patient users?
  - How user friendly is the platform?
  - Are staff comfortable with the display and type of data shown?
  - Which features are/are not useful to patients and clinicians?
  - Which features need removed or improved upon?
  - What, if any, bugs are encountered?
  - How accessible is the app/portal?
  - What is the optimal frequency of completing the patient log that is achievable and meaningful for asthma management?

2. **Process outcomes**: How does the implementation of AMAZE<sup>TM</sup> affect clinical process? For example, is patient communication improved, or is there an increase or decrease in time spent with patients?

The exploratory objectives are:

- 1. **Clinical outcomes**: How does the implementation of AMAZE<sup>TM</sup> affect clinical outcomes? For example, is there an increase or decrease in utilization of patient services, emergency department visits, or clinician contacts?
- 2. To identify which segments of patients are most likely to benefit from using AMAZE<sup>TM</sup>.

Since this study is exploratory regarding the feasibility, usability, and perceived benefit of using an electronic platform for disease management, there is no hypothesis testing.

#### **Methods:**

**Study design:** This is a longitudinal study in which the process of integrating the AMAZE<sup>TM</sup> disease management platform (DMP) into clinical practice will be assessed by implementing this program at MGH for six months.

For the clinical pilot study, patients with asthma of varying severity will be recruited. A target of up to 50 total patients will be recruited and consented for the purposes of the clinical pilot study, consisting of approximately 33 young adult (18-35 years old) and up to 17 adult patients (36 years of age and older). Approximate recruitment targets for the study include a subset of patients who are new to the practice (less than 3-month history with the practice) and with uncontrolled asthma (n = approx. 10) as well as patients experiencing at least 1 exacerbation in previous 12 months (n=approx. 40). Exacerbations are defined as a change in asthma symptoms requiring a course of oral steroids or steroid injection and/or a hospitalization or emergency department visit for asthma. MGH staff responsible for recruiting patients will participate in a training prior to recruitment starting, including the workflow for steps for the clinical pilot.

After collecting electronic informed consent via Research Electronic Data Capture (REDCap), participants will be instructed to download the AMAZE<sup>TM</sup> application software (app) to record their daily asthma symptoms and access educational materials and other features of the app. Participants will be allowed to retroactively complete their daily asthma symptoms log for up to 7 days prior to the current date. All entries will be date and time stamped to track entries. After downloading the app, participants will be emailed a sociodemographic form to complete. If the participant enables reminder notifications within the app, they will be sent one notification a day at their preferred time if they do not

access the app daily. On a monthly basis, the app will prompt them to complete the Asthma Control Test (ACT<sup>TM</sup>). Importantly, participant responses to the app will be monitored twice daily by a clinical and research team and alerts may be sent to their physician based on responses (e.g. participant reports of ED visits, multiple "bad" day reports, etc.) via the AMAZE<sup>TM</sup> interface to facilitate communication and to guide treatment.

A random selection of up to 12 participants will be asked to participate in longitudinal follow-up interviews at study months one, three, and six with the Evidera study team to monitor the implementation of the AMAZE<sup>TM</sup> platform. MGH personnel will be consented prior to completing any interviews. At study months 2, 4, and 5, a one-time random selection of up to 5 participants may be selected to complete a follow-up interview by the AZ DMP product team. During the follow-up longitudinal and cross-sectional interviews, participants will be asked questions regarding their use of the app/platform and what features may need improvements or are particularly of value.

Additionally, all participants will be asked to complete a patient user experience survey at study months 1, 3, and 6, as well as the System Usability Scale (SUS) at study months 1 and 6. All electronic surveys sent outside the app will be sent through REDCap. Clinical staff research participants will be asked to complete the SUS at study months one and six. Lastly, any time a participant attends a clinic visit (in-person or telehealth), they will be emailed a link to complete a patient visit experience satisfaction survey. At the end of the study, HCPs will be asked to complete a post-study survey via emailed link, while patients will be asked to complete the Patient Satisfaction Questionnaire (PSQ-18).

**Study Sites:** MGH outpatient adult and pediatric pulmonary clinics will be implementing the clinical pilot study.

**Data Source(s):** MGH was selected to implement AMAZE<sup>TM</sup> into their clinical practice based on the principal investigators' experience and qualifications, the number of asthma patients treated in the clinic, the diversity of the asthma patients treated by the clinic, the ability of the site to complete the study tasks in the allotted timeframe, and the anticipated unique component of clinical pilot initiatives anticipated by the study site.

**Study Population:** Clinic staff will invite eligible patients age ≥18 years with a diagnosis of asthma to enroll in the study. Up to 50 patients will be enrolled, including approximately 33 young adults (18-35 years old) and up to 17 adults (36 years of age and older).

#### **Exposure(s):**

Participants will complete the following measures at differing timepoints:

- AMAZE<sup>TM</sup> Patient App, including a daily symptom log, daily medications, healthcare resource utilization (HCRU), ACT<sup>TM</sup> completed every month, and educational resources
- Demographic characteristics questionnaire
- Patient User Experience Survey
- Patient Visit Experience Survey
- SUS
- Qualitative Semi-structured Interviews
- PSQ-18

MGH personnel will complete the following measures:

- Screening script for patient recruitment (CRC)
- Clinical Case Report Form (CRF) (CRC)
- Chart Review CRF (CRC)
- SUS (Clinical staff)
- Post-Study Survey (Clinical staff)

#### Outcome(s):

- Onboarding process evaluation
- Product attributes
- Patient visit and user experience
- Clinical staff experience
- Clinical process assessment
- SUS scores
- PSQ-18 scores
- Post-study survey responses
- Qualitative interview responses

**Sample Size Estimations:** As the aim of this study is to assess the process and feasibility of implementing AMAZE<sup>TM</sup>, inferential statistics will not be performed, and a formal sample size estimation is not applicable. MGH will target up to 50 patients. Implementing AMAZE<sup>TM</sup> among up to 50 patients will provide MGH with enough experience to provide feedback on the outcomes, barriers, benefits, challenges, ease of implementation, and areas for improvement for future integration as a platform.

**Statistical Analysis**: Descriptive statistics (n, frequency, mean, and standard deviation [SD]) will be used to characterize the sample in terms of sociodemographic and clinical characteristics. The sociodemographic and clinical characteristics will be summarized for the sample overall as well as for each site. Descriptive statistics (n, frequency, mean, and SD) will also be used to summarize the results from the patients' frequency of use of the daily log and educational resources, ACT<sup>TM</sup> scores, responses to the Patient Visit Experience Survey, the SUS, and the results of the patient PSQ-18 and HCP Post-study survey.

Qualitative interviews will be summarized based on interviewers' notes using a detailed interviewer matrix. The interviews will be audio recorded, and transcribed by a third-party vendor (TransPerfect), should the audio need to be reviewed to summarize findings. The interview results will be summarized in tabular format, with key recommendations, advantages, and disadvantages grouped. Specifically, barriers, benefits, challenges, ease of implementation, and areas for improvement will be summarized.

**Safety Handling Plan:** A Safety Handling Plan has not been developed for this study.

# **AMENDMENT HISTORY**

| Date | Section of study protocol | Amendment or update | Reason |
|------|---------------------------|---------------------|--------|
| | | N/A | |

# **MILESTONES**

| Milestone | Planned date |
|--------------------------------------|--------------|
| Final Protocol | Q4 2020 |
| Internal Review Board Approval | Q2 2021 |
| Site Trainings | Q2 2021 |
| First Participant In | Q2 2021 |
| Last Participant in | Q2 2021 |
| Database Lock | Q4 2021 |
| High Level Results in Tabular Format | Q4 2021 |
| Final Report | Q1 2022 |

#### 1. BACKGROUND AND RATIONALE

# 1.1 Background

Uncontrolled and severe uncontrolled asthma (SUA) are common disorders that are often difficult to identify and manage. The clinical and economic burden of SUA is disproportionately high, accounting for nearly 40% of asthma-related costs<sup>1,2</sup> and uncontrolled asthma affects over 50% of children and adults with asthma. With advances in asthma therapies, an urgent need exists to optimize uncontrolled and SUA recognition and clinical management.

#### 1.2 Rationale

Poor asthma control is often unrecognized as asthma patients learn to adapt to their disease and adjust to a suboptimal level of control. This can result in frequent exposure to systemic steroids along with frequent urgent care/ER visits and hospitalizations. The AMAZE<sup>TM</sup> platform aims to address this clinical need through better communication between patients and their clinical teams regarding the patients' level of asthma control with the ultimate goal of improvement asthma management and improved health outcomes. This study aims to test the feasibility of implementing AMAZE<sup>TM</sup> in a specialist clinical practice to manage asthma.

#### 2. OBJECTIVES AND HYPOTHESES

# 2.1 Primary Objective(s) and Hypothesis(es)

The primary study objective is to generate evidence on the feasibility, usability, perceived value, and potential benefits of the AMAZE<sup>TM</sup> disease management platform implemented in clinical practice. Since this is an exploratory study involving a mobile app and DMP, there is no hypothesis testing. The primary objective will be assessed through the following key outcomes:

- 1. **Technology Outcomes:** Key questions to be asked regarding the technology outcomes are:
  - How much is the platform utilized, and what is the perceived value by both clinical staff and patient users?
  - How user friendly is the platform?
  - Are staff comfortable with the display and type of data shown?
  - Which features are / are not useful to patients and clinicians?
  - Which features need removed or improved upon?
  - What if, any bugs, are encountered?

- How accessible is the app/portal?
- What is the optimal frequency of completing the patient log that is achievable and meaningful for asthma management?
- 2. **Process outcomes:** How does the implementation of AMAZE<sup>TM</sup> affect clinical process? For example, is patient communication improved, or is there an increase or decrease in time spent with patients?

# 2.2 Secondary Objective(s) and Hypothesis(es) (Optional)

There are no secondary objectives for this study.

# 2.3 Exploratory Objective(s) and Hypothesis(es) (Optional)

There are two exploratory objectives for this study.

- 1. **Clinical outcomes:** How does the implementation of AMAZE<sup>TM</sup> affect clinical outcomes? For example, is there an increase or decrease in utilization of patient services, emergency department visits, or clinician contacts?
- 2. To identify segments of patients that are most likely to benefit from using AMAZE<sup>TM</sup>.

#### 3. METHODOLOGY

# 3.1 Study Design – General Aspects

This is an implementation study to assess the feasibility, usability, perceived value, and potential benefits of integrating the AMAZE<sup>TM</sup> DMP at MGH. The AMAZE<sup>TM</sup> platform (developed by AstraZeneca/BrightInsight) consists of a clinician dashboard to guide treatment and asthma management, and a patient application to enter daily symptoms and medications that can trigger alerts to the clinician dashboard. For this implementation study, the sites will be trained on the use of the AMAZE<sup>TM</sup> platform and will launch the program in the target patient population.

For clinical pilot study launch, MGH will recruit up to 50 patients with asthma, including approximately 33 young adults (18–35 years old) and up to 17 adults. Approximately 10 new patients to the practice (less than 3-month history with the practice) but with uncontrolled asthma will be recruited, along with approximately 40 patients who have had at least one exacerbation per year. Eligible participants will be invited to participate in the study either in person or via telephone or Zoom call using a standardized recruitment script (Appendix A). Alternatively, a recruitment email will be first sent from a physician with a flyer attached to introduce the app and the study to participants (Appendix C). A follow-up Zoom video conversation can also be scheduled with the participants. If interested in participating in the study, they will provide their

email address to the site staff so that a consent form can be sent to them via email (Appendix B) to sign via REDCap. The MGH staff will confirm the email address provided by the participant is consistent with the email address within the DMP dashboard system. If the email address differs, the staff will modify the dashboard to the correct email. The email address collected during the screening visit will be used for emailing the surveys throughout the study. The MGH staff will review the consent with the patient either in person or via telephone or Zoom call and answer any questions they may have.

After consenting to participate, patients will be sent an introductory email (<u>Appendix D</u>) with link to download the app (<u>Appendix E</u>), and register as a patient with a unique identifier (ID). Once the app has been downloaded, the patient will be asked to create their unique ID. Within the app, participants will be provided with access to all educational materials and asked to complete the daily symptom log. The MGH research staff will complete a clinical case report form (CRF; <u>Appendix F</u>) to record baseline clinical information about the patient, while participants will be asked to complete a sociodemographic form (<u>Appendix G</u>) via an emailed link. If the participant enables reminder notifications within the app, they will be sent one notification a day at their preferred time if they do not complete the app daily. BreezoMeter, a third-party air quality vendor, will be assisting in the tracking and alerting of the air quality in the participant's location if the location setting is turned on.

After study launch, Evidera will conduct qualitative, longitudinal, follow-up interviews regarding process implementation with a random selection of patient participants (approximately 1 out of 5) at study months one, three, and six to gain a deeper understanding of the feasibility of implementing the asthma AMAZE<sup>TM</sup> platform. Prior to launching the interviews, approximately 12 patient participants will be randomly selected to participate in the qualitative interviews at study months one, three, and six to understand the feasibility and usability of the patient app over time, the perceived benefit (e.g., if there is an increase in the patient's ability to interact with their physician, if it enhances speed and/or quality of response, etc.), and how it can be improved. In addition to the longitudinal interviews, a one-time, cross-sectional interview may be conducted by the AZ DMP Product Team at months 2, 4, and 5 with a random selection of up to 5 patient participants at each timepoint (excluding the up to 12 participants who will be participating in the longitudinal interviews). The cross-sectional interviews are meant to help capture any new features or feedback from participants during the off-months in the longitudinal interviews and will be conducted on an as-needed basis.

In addition to the qualitative interviews, patient participants will be emailed a link to complete an electronic patient visit experience survey (<u>Appendix H</u>) after attending an in-person or telehealth visit with their doctor to evaluate their overall satisfaction with AMAZE<sup>TM</sup> and its impact on the visit. Evidera will receive a data report from BrightInsight with participant BrightInsight ID, date of visit, and status of visit completion. Evidera will then share the IDs with MGH to generate a

visit survey email. All participants will be asked to complete electronic Patient User Experience surveys, sent via email, as well as the SUS at study months one and six. These surveys are meant to allow participants the opportunity to provide feedback on the app as they continue to interact with the app longitudinally throughout the study. At the end of the study (approximately 3 months after completion of enrollment) prescribing providers and study coordinators at MGH will complete a Post-study Survey (Appendix I) and patient participants will complete the PSQ-18 (Appendix J). The focus of these questionnaires will be to obtain additional feedback on the implementation of AMAZE<sup>TM</sup> and participant satisfaction with the medical care they receive, respectively. All electronic surveys sent outside the app will be sent through REDCap. At study month Six, MGH staff will also be asked to complete a chart review CRF (Appendix K) for each patient. The patient app and/or clinician dashboard may be revised throughout the clinical pilot study based on feedback from patients and clinical staff.

#### 3.1.1 Data Source(s)

Participants will be recruited from MGH. MGH will recruit approximately 33 young adults (18–35 years old) and up to 17 adults for a total sample of up to 50 patients. In addition, MGH will aim to recruit patients who are new to the practice (less than 3-month history with the practice) but with uncontrolled asthma (n= approx. 10) and patients experiencing at least 1 exacerbation in previous 12 months (n=approx. 40).

# 3.2 Study Population

Clinic staff will invite patients age  $\ge 18$  years with an asthma diagnosis who are presenting for a clinic visit or via telephone to download the AMAZE<sup>TM</sup> App. Up to 50 patients will be recruited.

#### 3.3 Inclusion Criteria

Patients must meet all the following criteria to be considered for enrollment:

- 1.  $\geq$ 18 years of age at the time of enrollment
- 2. Clinically confirmed diagnosis of asthma (with or without COPD)
- 3. Access to a smartphone with internet access with the following requirements: iOS (Operating System iOS 13 or newer and Devices iPhone 8 or newer) or Android (Operating System 8.0 or newer)
- 4. Able to understand and speak English sufficiently to be able to use the AMAZE™ patient app
- 5. Willingness to participate in a telephone interview and be audio-recorded
- 6. Consenting to participate in the study

#### 3.4 Exclusion Criteria

Patients meeting any of the following criteria will not be included in the study:

- 1. No current diagnosis of asthma
- 2. Has a cognitive impairment, hearing difficulty, acute psychopathology, medical condition, or insufficient knowledge of the English language that, in the opinion of the investigator, would interfere with his or her ability to agree to participate and/or complete the ACT<sup>TM</sup>.

#### 4. VARIABLES AND EPIDEMIOLOGICAL MEASUREMENTS

## 4.1 Exposures

Prior to enrollment in the study, MGH staff will approach patients during an in-person or telehealth clinic visit or via telephone to assess interest and confirm eligibility. For the clinical study launch, a standardized screening script (Appendix A) will be used that provides an overview as to the purpose and nature of the implementation study, as well as a description of the potential to participate in the longitudinal or one-time follow-up interviews (if randomly selected to participate).

The timing of each key procedure/exposure, and the responsible party for each procedure is depicted below in Table 1. Following the baseline visit, Evidera will randomly select up to 12 patient participants for longitudinal interviews, as well as up to 5 participants per timepoint to take part in cross-sectional interviews. A detailed workflow of the implementation of the DMP in MGH clinical practice is included in <u>Appendix L</u>.

**Table 1. Schedule of Study Assessments** 

| Procedures | Baseline | Month<br>One | Month<br>Two | Month<br>Three | Month<br>Four | Month<br>Five | Month<br>Six |
|---|---|---|---|---|---|---|---|
| Screen and Recruit <sup>1</sup> | M | | | | | | |
| Consent via RedCap for Participants | M/P | | | | | | |
| Download App | P | | | | | | |
| Completion of App | P | P | P | P | P | P | P |
| Monitor Clinician<br>Dashboard | M | M | M | M | M | M | M |
| Clinical CRF | M | | | | | | |
| Sociodemographic Form | P | | | | | | |
| Patient User Experience<br>Survey | | P | | P | | | P |
| System Usability Scale | | P/M | | | | | P/M |

| Procedures | Baseline | Month<br>One | Month<br>Two | Month<br>Three | Month<br>Four | Month<br>Five | Month<br>Six |
|---|---|---|---|---|---|---|---|
| Patient Visit Experience<br>Survey <sup>2</sup> | | P | P | P | P | P | P |
| Participant Longitudinal Follow-up Interviews (n=approx. 12) | | P/E | | P/E | | | P/E |
| Participant Cross-sectional<br>Follow-up Interviews (n=<br>approx. 5) | | | P/AZ | | P/AZ | P/AZ | |
| Consent for MGH staff participating in surveys | | M | | | | | |
| Patient Satisfaction Questionnaire-18 | | | | | | | P |
| MGH Staff Post-Study<br>Survey | | | | | | | M |
| Chart Review CRF | | | | | | | M |

<sup>&</sup>lt;sup>1</sup>MGH will recruit approximately 50 patients for the clinical pilot study. Any additional patients invited to use the app beyond the maximum sample size will not be included in any analyses.

Abbreviation: AZ=AstraZeneca DMP Product Team; CRF = case report form; E=Evidera; M=MGH; P=Participant

Patient participants will be compensated \$10 after completion of applicable surveys from baseline through month 6. In addition, if a participant is randomly selected for an interview, they will also be compensated \$75 per interview completed. Patient participants will be randomized into one of three groups, and will only complete one of these groups:

- 1. Longitudinal (three total) interviews and receive up to \$265
- 2. Cross-sectional (one-time) interview and receive up to \$115
- 3. Not randomized to be interviewed and receive up to \$40

Below is a table outlining the remuneration payment schedule for patient participants.

**Table 2. Remuneration Payment Schedule for Patient Participants** 

| Procedures | Baseline | <b>Month One</b> | Month Three | Month Six |
|---|---|---|---|---|
| Completion of Electronic Surveys | \$10 | \$10 | \$10 | \$10 |
| Completion of Interview (if randomly selected) | | \$75 | \$75 | \$75 |
| <b>Total Possible Remuneration</b> | \$10 | \$85 | \$85 | \$85 |

<sup>&</sup>lt;sup>2</sup>The Patient Visit Experience Survey will be sent after a confirmed visit with their HCP at the site following baseline visit.

#### 4.1.1 Patient-Completed

### 4.1.1.1 AMAZE<sup>TM</sup> Patient App

At the initial baseline visit, participants will be asked to download the AMAZE<sup>TM</sup> app (Appendix D). The patient app includes a daily log of asthma symptoms, as well as additional questions on their asthma experience. As a part of the app, patients will have access to educational resources about their asthma and asthma medication. The resources are meant to be informative in nature based on how the participant responds to questions in their daily log. The app allows participants to communicate with the MGH staff as well as see daily and weekly trends in their asthma. My plan, a component within the app, contains medications, air quality and information regarding upcoming appointments.

Every four weeks, the ACT<sup>TM</sup> will also be administered and completed by the participant.<sup>3</sup> The ACT<sup>TM</sup> consists of five items with the total score used to identify participants with poor asthma control. The ACT<sup>TM</sup> classifies well controlled as  $\geq 20$ , not well controlled as 16–19, and very poorly controlled as  $\leq 15$ . The ACT<sup>TM</sup> questions with a four-week recall period address medication use, asthma symptoms and asthma-related impairment. The English version will be used in this study only.

#### 4.1.1.2 Patient Demographic Questionnaire

Participants will complete a brief self-administered Patient Demographic Questionnaire (Appendix G) following download of the patient application and providing their informed consent to participate; this questionnaire will be sent to all participating patients via an email link. This form collects the participant's age, ethnicity, living situation, employment, and education, and will be used to describe the sample and assist with interpreting the results.

#### 4.1.1.3 Patient User Experience Survey

All participants who consent to participate in the full clinical study will be emailed at months 1, 3, and 6 the patient user experience survey (Appendix M). The survey is meant to allow participants the opportunity to provide feedback on a monthly basis as they continue to interact with the app. The survey results will be reviewed to identify if any changes to the app are needed.

#### 4.1.1.4 Patient Visit Experience Survey

The patient visit experience survey (Appendix H) will be sent electronically any time a participant attends an in-person or telehealth clinic visit. Bright Insights will generate weekly reports to provide Evidera with IDs for those who completed clinic visits. Evidera will subsequently notify the electronic survey vendor to send the survey via email. This survey will evaluate patient satisfaction with their visit and any benefits the App provided for the visit.

#### 4.1.1.5 System Usability Scale

The System Usability Scale (SUS) (<u>Appendix N.1</u>) will be sent electronically at months one and six for participants to provide feedback on the AMAZE patient app. The SUS has been validated in previous usability studies to quantitatively evaluate the usability of a system, including mobile apps.<sup>4</sup>

#### 4.1.1.6 PSQ-18

At the end of the clinical pilot study (approximately 6 months), all participants who consented and participated in the clinical pilot study will be emailed a link to the Patient Satisfaction Questionnaire-18 (PSQ-18; <u>Appendix J</u>).<sup>5</sup> The PSQ-18 is a generic measure used to assess patient's overall satisfaction with their medical care and interactions with their HCPs. A higher score indicates greater satisfaction.

#### 4.1.1.7 Follow-up Process Interviews with Patients

#### **Longitudinal Interviews**

A semi-structured interview guide (<u>Appendix O</u>) will be used to obtain information from a randomly selected subset of patients at months one, three, and six during longitudinal, follow-up interviews to gain a deeper understanding of the feasibility of implementing the AMAZE<sup>TM</sup> platform. The semi-structured interview guides will include an introduction and follow with specific questions and probes designed to facilitate discussion and optimize consistency across interviews. The interview guide will elicit recommendations for improving the AMAZE platform experience for patients. Additional unscripted probes may also be used to gain further information or clarification. The interview guides may be modified as necessary during the study.

#### **Cross-Sectional Interviews**

Semi-structured interview guides for months 2, 4, and 5 (<u>Appendix O</u>) may be used to obtain information from a randomly selected subset of patients at months 2, 4, and 5 during one-time, follow-up interviews with the AZ DMP Product team to gain a deeper understanding of the usability of the AMAZE<sup>TM</sup> platform. The interviews will be conducted as needed. The interviews are meant to be briefly provide feedback on any new roll outs or issues with the app that cannot be captured during the longitudinal interviews. The semi-structured interview guides will include an introduction and follow with specific questions and probes designed to facilitate discussion and optimize consistency across interviews. The interview guide will elicit recommendations for improving the AMAZE platform experience for patients. Additional unscripted probes may also be used to gain further information or clarification. The interview guides may be modified as necessary during the study.

#### 4.1.2 MGH Completed

#### 4.1.2.1 Clinical Case Report Form

For each participant, MGH will complete a paper clinical case report form (CRF; <u>Appendix F</u>) during the initial site visit after informed consent is obtained. The clinical CRF serves to characterize patients based on their history of asthma, current medications, and the HCP's rating of the patient's asthma severity and control.

#### 4.1.2.2 Chart Review Case Report Form

For each participant, MGH will complete a chart review clinical CRF (<u>Appendix K</u>) at month six. The follow-up clinical CRF will evaluate exacerbation history during the last 6 months, healthcare resource utilization, change in therapy, and COVID-19 diagnosis.

### 4.1.2.3 System Usability Scale

The SUS (<u>Appendix N.2</u>) will be asked verbally to clinical staff during the telephone interviews at months one and six to provide feedback on the clinical dashboard.

#### 4.1.2.4 Post-study Survey

All clinical staff who participate will be asked to complete the Post-study Survey (<u>Appendix I</u>) after patient enrollment has completed (approximately four months after study launch). The purpose of this survey is to obtain feedback on the implementation of the AMAZE<sup>TM</sup> platform within each site's medical practice.

#### 4.2 Outcomes

#### 4.2.1 Primary Outcome

To address the primary objective to generate evidence on the feasibility, usability, perceived value, and potential benefits of the AMAZE<sup>TM</sup> implemented in clinical practice, the following outcomes will be assessed:

- Technology Outcomes: Technology outcomes will be assessed in a variety of ways throughout the clinical pilot study. Usage metrics will be collected by BrightInsight to assess the frequency of use by patients completing the daily log, and utilizing the educational resources provided. The usage of the clinical dashboard will also be tracked to evaluate the utility of the dashboard to MGH. Usage metrics will be analyzed by Evidera once provided by BrightInsight.
  - o The qualitative interviews from the longitudinal months one, three, and six interviews as well as the cross-sectional months two, four, and five interviews will provide data regarding the usefulness of the technology from a patient perspective.

- The patient user experience surveys may be evaluated as well to determine how the platform is being utilized and the user friendliness of the App.
- Process Outcomes: Similar to the technology outcomes described above, process outcomes will be evaluated using the patient follow-up interviews, patient visit experience survey, PSQ-18 scores, SUS scores, and post-study survey results. Analyses for the process outcomes will focus on variables evaluating the impact of AMAZE<sup>TM</sup> on clinical practice, including duration of patient visits and services, as well as responses to survey items on changes to timing of scheduling visits, communication during the visit, and satisfaction with medical care received.

#### 4.2.2 Secondary Outcome

There are no secondary objectives for this study.

#### **4.2.3 Exploratory Outcome One**

To address the first exploratory objective to assess how the implementation of AMAZE<sup>TM</sup> affects clinical outcomes, the following outcomes will be assessed:

• Clinical Outcomes: As part of AMAZE<sup>TM</sup>, all patients will be asked to utilize the App by completing the daily log and monthly ACT. Additionally, sites will be asked to complete a baseline clinical CRF and a six-month chart review CRF for each participant. The baseline clinical CRF will capture information on the patient's asthma and smoking history as well as current asthma medications. The chart review CRF will include questions on recent exacerbations, healthcare resource utilization, change in asthma therapy, and exposure to COVID-19. The variables collected from these CRFs will be used to evaluate how AMAZE<sup>TM</sup> impacts key clinical outcomes of interest. Descriptive statistics (n, frequency, mean, and SD) will be utilized.

#### 4.2.4 Exploratory Outcome Two

To address the second exploratory objective on identifying which segments of patients are most likely to benefit from using AMAZE<sup>TM</sup>, information collected from the patient sociodemographic form and clinical CRF will be used and analyses will be stratified by patient subgroups/segments. The following patient segments may be considered: age cohorts (TBD); sex; asthma severity cohorts (TBD); educational cohorts (TBD); and minority cohorts (TBD). Other patients' segments may be considered after reviewing sample distribution.

#### 4.3 Other Variables and Covariates

Demographic and/or clinical patient data will be used to summarize the sample overall and by site.

Study Protocol Form Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS\_001\_0016432824

#### 5. STATISTICAL ANALYSIS PLAN

## 5.1 Statistical Methods: General Aspects

Descriptive statistics (n, frequency, mean, and SD) will be used to characterize the sample in terms of sociodemographic and clinical characteristics. The sociodemographic and clinical characteristics will be summarized for the sample overall as well as for each site.

# 5.1.1 Primary Objective: To generate evidence on the feasibility, usability, perceived value, and potential benefits of the AMAZE<sup>TM</sup> implemented in clinical practice

The technology outcomes described in <u>section 4.2.1</u> above will be analyzed both qualitatively and quantitatively. The interview (longitudinal and cross-sectional follow-up) results will be summarized in tabular format, with key recommendations, advantages, and disadvantages grouped. Specifically, barriers, benefits, challenges, ease of implementation, and areas for improvement will be summarized. Results from the patient visit experience survey, monthly patient user experience surveys, PSQ-18, post-study survey, and usage metrics provided by BrightInsight will be analyzed using descriptive statistics (n, frequency, mean and SD).

The process outcomes described in <u>section 4.2.1</u> above will be analyzed similar to the technology outcomes. The interview results will be summarized in tabular format; survey results will be analyzed using descriptive statistics.

#### 5.1.2 Secondary Objective(s)

There are no secondary objectives for this study.

# 5.1.3 Exploratory Objective One: To assess how the implementation of AMAZE<sup>TM</sup> affects clinical outcomes

The variables collected from the baseline Clinical CRF and six-month chart review form will be used to evaluate how the AMAZE<sup>TM</sup> patient App impacts key clinical outcomes of interest (e.g. clinician visits, healthcare resource utilization, change in therapy). Descriptive statistics (n, frequency, mean, and SD) will be utilized.

# 5.1.4 Exploratory Objective Two: To identify patients who are most likely to benefit from using AMAZE<sup>TM</sup>

The variables collected form the patient sociodemographic form and Clinical CRF will be used to stratify patients into segments/subgroups. Proposed variables of interest are age, sex, asthma severity, educational subgroups, and minority status. Additional variables may also be used in the

exploratory analyses. Descriptive statistics (n, frequency, mean, and SD) will be used to characterize patients most likely to benefit from the App across these variables.

#### 5.2 Bias

#### 5.2.1 Methods to Minimize Bias

Bias may occur with patient selection into the study based on availability of the appropriate phone and operating system. For this initial implementation study, the age and sex of patients who are interested in participating but do not have access to the appropriate devices will be tracked.

#### 5.2.2 Adjustment for Multiple Comparisons

Not Applicable.

#### 5.2.3 Strengths and Limitations

The strengths of this study are that it aims to include a diverse sample of patients across MGH. The limitations of this study include that MGH may not be generalizable to all clinical sites treating asthma patients across the US and that the sample of patients may not be generalizable to all asthma patients ≥18 years of age.

## 5.3 Sample Size and Power Calculations

As the aim of this study is to assess the process and feasibility study of implementing the AMAZE<sup>TM</sup> in clinical practice, inferential statistics will not be conducted, and a formal sample size estimation is not applicable. MGH will target 50 patients. Implementing the AMAZE<sup>TM</sup> with up to 50 patients will provide MGH with enough experience to provide feedback on the outcomes, barriers, benefits, challenges, ease of implementation, and areas for improvement for future integration as a platform.

#### 6. STUDY CONDUCT AND REGULATORY DETAILS

# 6.1 Study Conduct

#### 6.1.1 Procedures

#### 6.1.1.1 Recruitment

Participants will be recruited from MGH. MGH will identify potential participants through chart/database/electronic medical record (EMR) reviews. Potentially eligible patients will also be identified using the Research Patient Data Registry (RDPR) Scheduled Query feature. We will search for patients diagnosed with asthma with or without COPD. Upon receipt of each updated patient list, study staff will perform a chart review of listed patients to confirm eligibility. Once patient eligibility is confirmed, study staff will provide the confirmed list to appropriate clinical

staff who, at their discretion, will approach their patients regarding participation in the research study.

MGH staff will approach patients during a regularly scheduled clinic visit or call potentially eligible participants and introduce the study using an introductory script (Appendix A). The script provides an overview as to the purpose and nature of each study. Alternatively, a recruitment email will be first sent from a physician with a flyer attached to introduce the app and the study to participants (Appendix C). A follow-up Zoom video conversation can also be scheduled with the participants. For the clinical pilot study, best efforts will be made to recruit approximately 10 patients who are new to the practice (less than 3-month history) but with uncontrolled asthma and approximately 40 patients experiencing at least 1 exacerbation in the previous 12 months. In addition, over half the sample will be young adults (18–35 years old). The research staff will document patient interest and the recruitment quota using the Recruitment Tracking Log (Appendix P), including documentation of the number of patients who choose not to participate.

#### **6.1.1.2** Baseline Visit

During the baseline visit, interested participants that have verbally consented to participate will be sent an email (Appendix B) by the clinic staff via REDCap to provide electronic consent to participate in the clinical pilot study. The email address will be confirmed during screening and staff will add the email address in the dashboard system if it differs from the email address in the dashboard. MGH staff will review the consent either in person or via telephone and answer any questions they may have. Once the participant and MGH staff have signed, a fully executed version will be available for download. The consent will acknowledge the random selection of patients who will be asked to complete either a longitudinal or cross-sectional follow-up interview. After consent, patients will be provided with a link to download the App (Appendix E) and register as a patient with a unique identifier (ID). After completion of the baseline visit, patients will be emailed a brief sociodemographic questionnaire (Appendix G). MGH will also be asked to complete a clinical CRF (Appendix F) to capture initial clinical characteristics. Patients will be remunerated \$10 for completing the sociodemographic questionnaire at the baseline visit. Evidera will provide the email addresses collected at the screening visit to the web survey vendor in order to email the follow-up survey links.

#### 6.1.1.3 Longitudinal Follow-up Interviews and Assessments

Throughout the study duration, participants will be able to access the daily log of symptoms, questions on their asthma experience, and educational resources each day they interact with the AMAZE<sup>TM</sup> app. Every month, the app will prompt the completion of the ACT<sup>TM</sup>. Based on the responses on the patient App, a notification or alert may be triggered in the clinician dashboard for the sites to contact the patient and assess the severity of their symptoms and propose next steps (e.g., complete a clinic visit). In addition to the daily App completion, patients will be emailed a

monthly patient user survey to complete, as well as the SUS at months one and six. Patients will be remunerated \$10 with payment at months 1, 3, and 6 on their ClinCard for completion of applicable surveys. In addition, patients who are randomly selected will be compensated \$75 for each successfully completed interview.

Up to 12 randomly selected patients from MGH will be asked to participate in qualitative, longitudinal, follow-up interviews at months one, three, and six to evaluate the implementation and convenience of AMAZE<sup>TM</sup>. Interviews will be conducted over the phone with Evidera staff. The interviews will be audio recorded and transcribed by a third-party vendor (TransPerfect). Interviews are expected to last approximately 30 to 45 minutes for patients. Patients will be remunerated \$75 for their time via ClinCard at each interview time point.

#### 6.1.1.4 Cross-Sectional Follow-up Interviews and Assessments

Participants will be asked to complete the patient visit experience survey after attending an inperson or telehealth visit with their doctor. The survey will be emailed to participants after confirmation of completion of the visit.

A random selection of up to 5 patients at MGH will be asked to participate in a cross-sectional, one-time, follow-up interview either at month two, four, or five. The cross-sectional interviews will be conducted by AZ DMP Product team. Evidera will contact the participants to schedule the cross-sectional interview. To maintain data privacy, a teleconference line will be provided to the participants and AZ team. The goal of the one-time interview will be to evaluate any usability and feasibility issues with patients and provide an opportunity for participants to provide feedback on areas for growth or change in the patient App that cannot be captured during longitudinal interviews. Patient participants will be remunerated \$75 at the completion of the interview and paid at months 2, 4, and 5.

Approximately 6 months after first patient in, MGH staff will be asked to complete a post-study survey and patients will complete the PSQ-18, both provided via email to provide final feedback on the implementation of feasibility of the AMAZE<sup>TM</sup> patient App and clinician dashboard, and satisfaction with medical care received, respectively. MGH staff will also complete a 6-month clinical CRF.

#### 6.1.1.5 Claims Data Export

After the participants consent to participate, Evidera, and AZ will work to export deidentified claims data at months 6. The linking of deidentified data with the clinical pilot de-identified data will be outlined in detail in a subsequent study amendment prior to month 3. Alternatively, claims data may be linked to clinical pilot participants. The processes related to claims linking will be revised during an amendment. Any procedures related to this will not be implemented until IRB approved.

Study Protocol Form Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS\_001\_0016432828

### **6.1.2 Quality Control**

#### 6.1.2.1 Monitoring

Before the first subject is recruited into the study, the Medical Evidence and Observational Research (MEOR) Delivery Director, MEOR Operations Lead or CRO Representative (i.e., Evidera) will:

- Establish the adequacy of the facilities and the investigator's capability to appropriately select the sample; and
- Discuss with the investigator(s) (and other personnel involved with the study) their
  responsibilities with regards to protocol compliance, and the responsibilities of AZ or its
  representatives. This will be documented in an Interventional Study Primary Agreement or
  equivalent between AZ/delegate and the investigator.

During the study the local marketing company (MC) representative or delegate can implement different activities to assure compliance with AZ standards of quality. These activities could include but are not limited to:

#### 6.1.2.2 Contacts with the sites to:

- Provide information and support to the investigator(s)
- Confirm that the research team is complying with the protocol and that data are being accurately recorded in the CRFs
- Ensure that the CRFs are completed properly and with adequate quality

#### **6.1.2.3** Remote Monitoring activities for:

- Checking informed consent forms (ICF)
- Review enrollment forms and subsequent CRFs
- Export of claims data

The extent and nature of monitoring will be decided during the study planning based on design, complexity, number of subjects, number of sites, etc. Interventional Research Center (multi country)/MC will give some recommendations that could be locally adapted.

Different signals (e.g., high rejection rate in a site) should be used as potential identification of low protocol compliance by investigators.

If these or any other signal occurs or if the CRO is suspicious of a potential non-optimal level of protocol compliance by the site investigator, specific measures should be adopted to evaluate the situation, identify the issue and implement specific action plans to correct the situation.

# 6.1.2.4 Training of Study Site Personnel

Evidera will ensure training of MGH personnel for the implementation of AMAZE<sup>TM</sup> clinical pilot study procedures outlined in the study protocol. MGH principal investigators will ensure that appropriate training relevant to the study is provided to MGH staff, and that any new information relevant to the performance of this study is forwarded to the staff involved.

#### 6.1.2.5 ePRO Programming and Hosting

REDCap will be used for the electronic patient and clinical site staff surveys and clinical case report forms (CRFs). The survey hosted will include the sociodemographic form, monthly patient user experience survey, patient visit experience survey, SUS, post-study survey, and PSQ-18. A separate HIPAA-compliant vendor, BrightInsight, will host the data management system to collect and monitor data captured by AMAZE<sup>TM</sup>.

For both vendors, the quality assurance process will include extensive end-to-end testing. During all data collection, the survey responses will be tracked by unique participant identifiers—not participant names. All electronic surveys will be emailed to patient participants and clinical staff research participant through REDCap.

MGH will export and transfer the CRF and survey data in SAS format to Evidera via MGB Secure File Transfer. The CRF and survey data will then be entered into the database and reviewed by project scientific staff. Data discrepancies will be identified and resolved.

The web survey developed for the patient and MGH staff surveys will be tested prior to study launch.

# 6.2 Protection of Human Subjects

This Interventional Study will be performed in accordance with ethical principles that are consistent with the Declaration of Helsinki, ICH GCPs, GPP and the applicable legislation on Non-Interventional Studies and/or Interventional Studies.

The Investigator will perform the clinical pilot Study in accordance with the regulations and guidelines governing medical practice and ethics in the country of the clinical pilot Study and in accordance with currently acceptable techniques and know-how.

The final protocol of the clinical pilot Study, including the final version of the Patient Informed Consent Form, must be approved or given a favourable opinion in writing by the Ethics Committee/Institutional Review Board (IRB)/Independent Ethics Committee (IEC).

The Ethics Committee/IRB/IEC must also approve any amendment to the protocol and all advertising used to recruit subjects for the study, according to local regulations.

#### 6.2.1 Informed Consent

MGH staff will be responsible for ensuring that each participant (patients and MGH staff) fully understands the study's nature, purpose, procedures, risks, and benefits. For those patients and MGH staff taking part in the clinical pilot launch, electronic consent will be presented to them via REDCap. At the screening, the MGH staff will confirm the email address to send the REDCap document to and update the dashboard as needed with any patient email addresses that are not in the system. Evidera will provide the email addresses collected at the baseline visit to the webbased survey vendor via secure portal. MGH staff will review the consent (either in person or via telephone) and answer any questions. MGH staff will confirm the email address with the participant during the initial screening process.

Participants (patients and MGH staff) will also be informed of their rights as a participant, including that they may refuse to take part or withdraw at any time without penalty or giving up any benefits to which they are otherwise entitled. The participants also will be informed that, should they choose not to participate in all or any part of the study, their current or future treatment at the site will not be affected.

This study involves participant-completed measures for information purposes only; the study does not involve the use of an investigational drug or device. There are no known risks or benefits to participants. During or following the research study, patients may become more aware of how they feel about their condition—and how their condition may affect certain aspects of their life. Patients will be encouraged to talk with their asthma provider about their questions or concerns. The elements of federal regulations pertaining to consent procedures, disclosure of potential risks and benefits, and patient confidentiality will be strictly observed.

#### 6.2.2 Confidentiality of Study/Patient Data

All data collected will be strictly confidential, in accordance with local, state, and federal law. Personnel from the following organizations may examine the research study records: Evidera, AZ, and regulatory agencies (such as the FDA and the IRB). Only MGH staff involved in participant recruitment, clinical data extraction, and questionnaire administration will know the identities of the patients. Staff will be instructed to maintain complete confidentiality of all collected data. Participant data files collected by MGH and shared with either Evidera or AZ will be kept in a locked file cabinet separate from their identifying information and will be destroyed per Evidera's SOPs after a period of seven years. The summary report generated from the completed questionnaires will not contain any participant-identifying information. Medical data collected will not be associated with personal health identification data. All study data will be de-identified.

Evidera retains records for a minimum of two years on site, and an additional five years off site. Upon enrollment, participants will be assigned unique identification numbers. These unique

identifiers will be used to track the participants throughout the study. Only the unique participant identification numbers and participant initials will be entered into the database and recorded on the participant questionnaires—not participant names.

This interventional study will be performed in accordance with ethical principles that are consistent with the Declaration of Helsinki, International Council for Harmonization (ICH), Good Clinical Practice (GCP), and the applicable legislation on Interventional Studies.

The investigators will perform the clinical pilot study in accordance with the regulations and guidelines governing medical practice and ethics in the country of the interventional study, and in accordance with currently acceptable techniques and know-how.

The final clinical pilot study protocol, including the final version of the Patient and MGH Informed Consent Form, must be approved or given a favorable opinion in writing by the Ethics Committee/IRB/Independent Ethics Committee (IEC).

The Ethics Committee/IRB/IEC must also approve any protocol amendment and all advertising used to recruit subjects for the study, according to local regulations.

### 6.3 Collection and Reporting of Adverse Events/Adverse Drug Reactions

#### 6.3.1 Collection of Adverse Events

This is an interventional study with no requirements to actively collect adverse events during the study since enrollment in the study is based on disease diagnosis and does not require the administration of an AZ drug. However, if an investigator (or patient) would like to report an AE that is not required to be collected, this can be reported as a spontaneous report according to local regulations. The open-ended question in the feedback section of the App will be monitored for AE reporting by the AZ Production team.

#### **6.3.2** Reporting of Adverse Events

It is not necessary to report potential AEs based on answers to the ACT<sup>TM</sup>.

The rationale is, the signs and symptoms collected by these instruments are prevalent among asthmatic patients. It is not feasible to evaluate associations between a specific drug and events reported by patients based on these instruments due to lack of baseline disease information and temporal relationship of drug and event. According to the literature, more than 50% of asthma patients who are under medication will have such signs and symptoms.

Patients will be informed that their healthcare providers (including MGH staff and their clinician) will not be reviewing their responses to the study questionnaires in real time. They will be

instructed to report any health concerns or issues that they may experience directly to their healthcare providers.

#### 6.3.3 Aggregate Safety Review from PRO Instruments

An aggregate data report (in the form of a summary) of the PROs' scores from patients on AZ product(s) will be provided to the Global Safety Physician (GSP) and Safety Surveillance and Management Team (SSaMT) Lead for their review at the end of the study, so that the data can be considered in the context of the overall benefit: risk assessment of the product(s).

### 7. REFERENCES

- 1. Moore WC, Bleecker ER, Curran-Everett D, et al. Characterization of the severe asthma phenotype by the National Heart, Lung, and Blood Institute's Severe Asthma Research Program. *J Allergy Clin Immunol*. 2007;119(2):405-413.
- 2. Nunes C, Pereira AM, Morais-Almeida M. Asthma costs and social impact. *Asthma Research and Practice*. 2017;3(1):1.
- 3. Nathan RA, Sorkness CA, Kosinski M, et al. Development of the asthma control test: a survey for assessing asthma control. *J Allergy Clin Immunol*. 2004;113(1):59-65.
- 4. Bangor A, Kortum PT, Miller JT. An Empirical Evaluation of the System Usability Scale. *International Journal of Human–Computer Interaction*. 2008;24(6):574-594.
- 5. Marshall GN HR. The Patient Satisfaction Questionnaire Short-Form (PSQ-18). In. Santa Monica, CA: Rand Corp.; 1994.

#### 8. APPENDIX A. PATIENT SCREENING SCRIPT

Prior to initiating screening contact, please confirm the following from the patient's chart:

| The patient has a clinical diagnosis of asthma | Confirmed □ |
|---|---|
| The patient is at least 18 years of age (Recruitment quota: approximately 33 young adult patients (18–35 years of age) | Confirmed □ |
| Recruitment Quota only: New patients to the practice (less than 3-month history) and with uncontrolled asthma | Confirmed □ |
| Recruitment Quota only: At least one exacerbation per year | Confirmed □ |

#### **Introductory Script for Clinical Pilot Study Participants**

| Hello [patient name], my name is [interviewer name] and I am working with MGH and |
|---|
| AstraZeneca on a research study to evaluate a new smart phone app called AMAZE <sup>TM</sup> to monitor |
| asthma symptoms and to provide resources that may be helpful for asthma patients like you. I will |
| provide some basic information about this study and ask you some questions to find out if you |
| might qualify for the study. This conversation will take about 20 minutes, is this a good time to |
| talk?Yes No |

If no, thank you for your time today!

If yes, thank you for your interest.

We are participating in a research study with Evidera and AstraZeneca, a health outcomes research organization and Pharmaceutical company, to evaluate a new patient App that will help you monitor your asthma daily and provide resources that may be helpful for asthma patients like you. The goal of this study is to see if the patient App helps improve your care. Information from your medical records, such as your age, medications, existing medical conditions, will be collected for this study.

You will be asked to use the App over the next six months by completing the daily questions and will have access to educational materials provided in the App. A brief sociodemographic form will be sent via email for your completion, as well as periodic surveys to gain additional

information about your experiences using the App. If you agree to participate, you will be emailed a link to download the App with a unique ID. You will be compensated \$10 for each visit completed and paid at baseline, months 1, 3 and 6 for a potential total of \$40.

As a part of this study, some participants will be randomly selected to complete a series of telephone interviews (around 1, 3, and 6 months after enrolling in the study) or just one interview (around 2, 4, or 5 months after enrolling in the study) to be conducted by Evidera or AstraZeneca. If selected for the interviews, the interview will be audio recorded and transcribed by a third-party vendor (TransPerfect), and should last approximately 30 to 45 minutes.

Subjects will get \$10 for each visit completed and \$75 for each interview. The maximum each subject may receive for completion of visits is \$40. Subjects will be randomized into one of three groups. Participants will only complete one of these groups:

- 4. Longitudinal (three total) interviews and receive up to \$265
- 5. Cross-sectional (one-time) interviews and receive up to \$115
- 6. Not randomized to be interviewed and receive up to \$40

As a participant in this research study, there will be no direct benefits for you; however, information from this study may help health care providers improve the way they ask patients questions about their asthma.

The risks of the study are expected to be minimal. There is the risk that allowing us to record your name with your answers and accessing your health information is a possible loss of confidentiality. We will take reasonable steps to protect the confidentiality of your information.

Taking part in this study is voluntary. You may choose not to take part in this study, or if you decide to take part, you can change your mind later and withdraw from the study. Your decision will not change any present or future relationships with MGH or its affiliates.

| Are you interested in participating this study?YesNo |
|---|
| If no, thank you for your time today! |
| If yes, thank you for your interest. |
| Before moving forward, would you be willing to answer some questions to find out if you might qualify for the study? I will record your answers in writing, but only collect detailed contact information if you qualify for the study. May I begin? Yes No |
| Can you confirm if you have a smartphone with internet access?YesNo |
|---|
| If yes, what type of smartphone and operating system do you have?iPhone (OS and Type) Android (OS)Other |
| If the participant does not have an iPhone 8 or newer with an Operating System of 13 or newer or an Android with an Operating System of 8.0 or newer, the participant is not eligible to participate and thank them for their time! |
| As a part of the study you will be sent an emailed link with your unique ID to log-in to the application as well as instructions for how to download the app. |
| I need to collect some information from you to share with Evidera in order to make your profile for the reloadable gift card, ClinCard, and share your email address for sending you the study consent form and for future survey completion. |
| Do you grant permission for the study team to send you the full study consent form via email for you to review and sign?YesNo |
| Do you grant permission for the study team to leave a brief voice mail message if you are not available when the study team schedules calls? Yes No |

## Contact Information (AMAZE<sup>TM</sup> App)

Dear Research Participant,

Thank you for taking part of the AMAZE<sup>TM</sup> Asthma Research Study at Massachusetts General Hospital (MGH).

As part of the study procedure, please complete the form below to confirm your contact information. This will be used to set up your profile for payment.

| If you have any questions, please | contact the Study Te | eam at <mark>CC</mark> I | |
|---|---|---|---|
| Thank you! | | | |
| First Name (Please enter your Fir initial) | | ot use an | |
| Last Name (Please enter your Lasinitial) | st Name in full, do no | ot use an | |
| Date of birth: | | | |
| Street or PO Address: | | | |
| City: | State: | Zip code: | |
| Phone Number: (Home) | (Work) | (Cell) | |
| Email: | | | |
| Do you grant permission for the savailable when the study team solution and the study team solution to the savailable when the study team solution to the savailable when the study team solution to the savailable when the savailable when the savailab | hedules calls? | brief voice mail message if you a | ire not |
| Best time to call (Monday-Friday | 9am-5pm): | | |

#### APPENDIX B. ELECTRONIC CONSENT EMAIL 9.

### **Signature Line Subject:**

AMAZE<sup>TM</sup> Health Management MGH Asthma Mobile App Study – Electronic Consent Form



#### 10. APPENDIX C. RECRUITMENT EMAIL AND FLYER

#### Recruitment email to be sent to the patient participants:

**Subject**: MGH AMAZE Asthma Study Participation **Attach**: MGH Flyer PDF (**check latest version of this**)

Dear Salutation Last Name,

We invite you to participate in a research study alongside AstraZeneca (a pharmaceutical company) and Evidera (a health outcomes research organization) to evaluate a smartphone application (app) called, AMAZE<sup>TM</sup> that may assist you in monitoring your asthma on a daily basis. The overall goal of this study is to evaluate if the patient App helps improves your care!

If interested, and you decide to participate in this voluntary study, you will be asked to use the App for six months by completing a daily assessment logs (~1 minute per day). You will also be asked to complete periodic user feedback surveys to gain insight about your experiences using the App. There will be total of approximately 7 surveys throughout the study and would take no more than a few minutes to complete each, and you would receive \$40 total for completion of all surveys. For this study, if you choose to participate, some participants will also be asked to be randomly selected to complete a set of three telephone interviews (or a one-time interview) which will be conducted by Evidera, our health outcomes collaborator. For these additional interviews, you will be paid \$75 for each completed interview (if randomly selected).

The risks of the study are expected to be minimal. There is the risk that allowing us to record your name with your answers and accessing your health information is a possible loss of confidentiality. We will take reasonable steps to protect the confidentiality of all your information.

If you are interested, please respond to this email and we can set up a brief discussion to address project details and the informed consent documentation. Following the informed consent process, we can then download the app and set up your account.

Attached is the study flyer providing a brief introduction to the app.

We look forward to your response either way!

Thanks in advance,

Signature block of provider and either PPD

or PPD

MGH AMAZE<sup>TM</sup> Asthma Study Team Massachusetts General Hospital 55 Fruit St. Boston, MA 02114

CCI

## Recruitment email to be sent to the clinical staff research participant:

| Dear |
|---|
| Thank you for your interest in our research study about a newly developed mobile app for asthma patients. In this research study we want to evaluate the AMAZE <sup>TM</sup> App to help monitor MGH asthma patients. The goal of this study is to learn about the impact of this digital disease management platform on the quality of life, outcomes, and treatment of asthma patients. |
| If you decide to join this research study, it will take you about 6 months to complete the study. You will be asked to provide your personal opinion (by completing the post-study survey and system usability scale surveys), as a MGH clinical staff involved in the study, to gain a deeper understanding of the feasibility of implementing the asthma AMAZE <sup>TM</sup> platform. There will be a total of 3 surveys throughout the research study and would take no more than a few minutes to complete each survey, and you will not be paid for completing these surveys. |
| Prior to participating in the study, you will need to provide consent electronically. When invited to do so by the study staff, please go to the following URL: <insert consent="" url=""></insert> |
| For questions, please send an email to the study team: CCI |
| Thanks, |
| MGH AMAZE <sup>TM</sup> Asthma Study Team |



## A research study to monitor your asthma through an app:

## **Introducing Key Features**



#### **Daily Log**

Share information like symptoms, triggers, and more directly with your care team.



#### **Trends**

Spot patterns in your asthma through weekly charts and graphs.



#### Medications

View your list of medications and set reminders so you never forget to take them.



#### **Air Quality**

See the latest air quality conditions and set air alerts so you know when it is safe out.



#### Messaging

Message your care team any non-urgent medical questions.



#### Safe and Secure

Your personally identified health data will be safe and secure on the platform and only shared directly with your care team.



#### **Amaze App**

Stay connected for better asthma control







If you have any questions, please contact the research study team at:



#### 11. APPENDIX D. INTRODUCTORY EMAIL

The code and invitation code expiration date and time will be modified for each individual participant.



#### Welcome to Mass General Hospital

It is our pleasure to offer you a free app to help you track your asthma symptoms, communicate with your care team, monitor air quality, and much more.

It only takes a moment to setup:

1. Download the app to your device





- 2. Create an account
- 3. When prompted for an invitation code, enter the code below:

098639

4. Start logging your symptoms

Your invitation code expires on 08/19/2020 at 3:04 PM

The invitation code is unique to the patient who received the code in their email - please do not share it. Data entered in the app will be associated with the patient who received the invitation code.

# 12. APPENDIX E. AMAZE<sup>TM</sup> PATIENT MOBILE APPLICATION SCREENSHOTS

## 12.1 Flyer for App







Study Protocol Form Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS 001 0016432844

Messaging

medical questions.

Safe and Secure

Message your care team any non-urgent

Your personally identified health data will be safe and secure on the platform and only shared directly with your care team.

## 12.2 Account Creation and Login

9:41



# Welcome to Massachusetts General Hospital



## Keep your doctor updated.

Track your health in your log each day so your doctor knows how you are doing.



## Better understand your health.

Review your week to spot patterns between symptoms, triggers, medication use, and more.



## Share your data to help others.

Share your anonymous data to help healthcare providers better understand chronic conditions to help people like you.

Next



## 9:41

## .ul 중 🗩

## Add phone number

#### Mobile Phone Number

Required

Continue



## Let's begin your first log!

Track your health in your log each day so your doctor stays updated on how you are doing.

**Begin Daily Log** 

**Date August 10, 2021** 

No SIM 🕏

10:02 AM



## Welcome to **Massachusetts General** Hospital



Take control of your health.

#### Create an account

Login

Manufactured by BrightInsight Inc. Version 1.1



## **Email verification code**

This 6-digit code has been sent to the email you provided.

Verify



## Welcome!

Your account has been successfully created.

**Get Started** 

Didn't receive the code? Tap here

## 12.3 Terms of Use



AZ - MGH - AMAZE DMP - Clinician Port

Study Protocol Form Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS\_001\_0016432849



AZ - MGH - AMAZE DMP - Privacy Policy



AZ - MGH - AMAZE DMP - Patient Terms

## 12.4 Air Quality





Study Protocol Form Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS 001 0016432851

| 9:41 | | .il 중 🔳 |
|------------|-------|-----------------|
| Cancel | Trees | |
| Pine | | None |
| Juniper | | Very high - 5/5 |
| Elm | | Off season |
| Oak | | High - 4/5 |
| Alder | | Off season |
| Cottonwood | | Off season |
| Birch | | Off season |
| Ash | | Off season |
| Maple | | Off season |

| 9:41 | | .ıl ≎ ■ |
|-------------|-------------|------------|
| | Pollen Info | Close |
| Score range | | |
| Very Low | | 1 out of 5 |
| Low | | 2 out of 5 |
| Moderate | | 3 out of 5 |
| High | | 4 out of 5 |
| Very High | | 5 out of 5 |
| D. II | | |

Pollen is a common allergen that can cause an allergic asthma. A pollen count is a measure of the concentration of all the pollen in the air in a certain area at a specific time.

The severity levels above (very low to very high) is based on various parameters that predict the probable allergic symptoms intensity.

If pollen is an asthma trigger for you, you can reduce your exposure to pollen by:

- Limiting outdoor activities when pollen is high.
- Consider an activated air filtration system.
- Keeping windows closed during pollen season.
- Wear sunglasses and a hat outdoors.
- Changing and washing clothes after being outside.

Also, keep an eye on your local weather: dry, windy, sunny days drive higher pollen counts while rain, moisture, and cloudy conditions generally keep pollen numbers down.



Breathing in humid air activates nerves in your lungs that narrow and tighten your airways.

Humidity also makes the air stagnant enough to trap pollutants and allergens like pollen, dust, mold, dust mites, and smoke. These can set off your asthma symptoms.

Humidity over 60 percent also encourages the growth of mold. If you're sensitive to mold, breathing it in can flare up your asthma.

Dust mites live in furniture, carpets, and bedding. They thrive at humidity levels of 70 to 80 percent. Their dead bodies and waste can also set off asthma attacks.

## 12.5 Appointments

Study Protocol Form Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS\_001\_0016432853

#### 12.6 Asthma Control Test

## Asthma Control Test™

© QualityMetric Incorporated 2002, 2004, 2011. All rights reserved.

Asthma Control Test™ is a trademark of QualityMetric Incorporated.

United States (English) version.

Next



## Asthma Control Test™

This survey was designed to help you describe your asthma and how your asthma affects how you feel and what you are able to do. For each of the following questions, please select the one response that best describes your answer.

Next

Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4

**Date August 10, 2021** 



During the <u>past 4 weeks</u>, how often did your <u>asthma</u> symptoms (wheezing, coughing, shortness of breath, chest tightness or pain) wake you at night or earlier than usual in the morning?



#### Date August 10, 2021





Previous

Next

**Previous** 

Save

## 12.7 Daily Asthma Log



# Have you taken any of these medications for asthma today?

## Maintenance / daily No Taken every day to maintain control of your asthma (e.g., Flovent, Symbicort, Advair, etc.). This would also include rescue medication (e.g., albuterol) that you take on a regular basis for exercise. Oral steroids (i.e., prednisone) Taken for a short period of time if/when your No asthma symptoms worsen. If you take oral steroids every day either for your asthma or another condition, do NOT include that here. Quick-relief / as-needed No Taken only when you experience symptoms of your asthma. If you regularly use rescue medication prior to exercise, select the "maintenance" option instead. **Previous** Next

Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4

#### Date August 10, 2021



Version 7.4 Form Doc ID: AZDoc0059948

Parent Doc ID: SOP LDMS\_001\_0016432860



## How do you feel today?

Tap on a face below (required)





Good

**Next** 



Version 7.4
Form Doc ID: AZDoc0059948
Parent Doc ID: SOP LDMS 001 0016432861





**Previous** 

**Next** 



### Call 911 for medical emergency!

If you think you are experiencing a medical emergency, get directions to the nearest hospital or call 911.

# Call 911

Call emergency help directly from the app

#### Seach nearby hospitals

Get directions to a nearby emergency room by launching your device's map app

I'm okay, proceed!



## Version 7.4 **Date August 10, 2021**



Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4

#### **Date August 10, 2021**



Version 7.4

Form Doc ID: AZDoc0059948

Parent Doc ID: SOP LDMS\_001\_0016432865

#### **Date August 10, 2021**

## 12.8 Education

No SIM 🗢

10:07 AM

@ 1 1

< Home

Education



#### The basics of asthma

Learn the basics of asthma and explore resources from the CDC about better controlling your asthma.



#### Diagnosing asthma

Understand how asthma is diagnosed and the different types of tests involved.



#### Common asthma triggers

Explore the most common asthma triggers from tobacco smoke to air pollution to pets and how you should avoid them.



#### Asthma action plan

Understand what an asthma action plan is and why they are important as well as a link to one you can create with your doctor.



#### Asthma resources and videos

Explore resources and videos on how to use your inhaler correctly, pursed lip breathing, and using a peak flow meter.



## Symptoms, causes and risk factors

Know how to recognize common asthma symptoms and what you can do about them along with asthma causes and risk factors.



## Asthma Treatment and Management

Learn how asthma is commonly treated and controlled and how you can try and prevent attacks.



#### Controlling your asthma

Better understand what causes asthma attacks and how to recognize them as well as how to gain better control of your asthma.



#### Living with asthma

Find support and tips on how you can best live with your asthma and still be as active and as healthy as possible.



#### Asthma online support group

Check out Inspire, the asthma support and discussion community where you can connect with others living with asthma.











Study Protocol Form Version 7.4

Form Doc ID: AZDoc0059948

Parent Doc ID: SOP LDMS 001 0016432866

## 12.9 Email Password Reset

#### 12.10 Home





#### Your Care Team's Request





Study Protocol Form Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS\_001\_0016432868

## 12.11 Messages

## Messages



Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4

**Date August 10, 2021** 



| ◆ TestFlight ◆ | 3:23 PM | @ <b>1</b> |
|------------------|------------------|------------|
| <b>&lt;</b> Back | Choose Subject | |
| Non-urgent n | nedical question | 0 |
| Prescription o | question | $\circ$ |
| Test results q | uestion | $\circ$ |
| Visit follow-u | o question | $\circ$ |
| Referral requ | est | $\bigcirc$ |

Disclaimer: Messages are not for medical emergencies. For medical emergencies, call 911 immediately.

### Messages



#### 12.12 Feedback


### **12.13** My Plan



#### **Budesonide Oral Inhalation**

Budesonide is used to prevent difficulty breathing, chest tightness, wheezing, and coughing caused by asthma. Budesonide powder for oral inhalation (Pulmicort Flexhaler) is used in adults and children 6 years of age and older. Budesonide suspension (liquid) for oral inhalation (Pulmicort Respules) is used in children 12 months to 8 years of age. Budesonide belongs to a class of medications called corticosteroids. It works by decreasing swelling and irritation in the airways to allow for easier breathing.

Learn More

#### Formoterol oral inhalation

Formoterol oral inhalation is used to control wheezing, shortness of breath, and chest tightness caused by chronic obstructive pulmonary disease (COPD; a group of lung diseases that includes chronic bronchitis and emphysema). Formoterol is in a class of medications called long-acting beta agonists (LABAs). It works by relaxing and opening air passages in the lungs, making it easier to breathe.

Learn More

FORMOTEROL)



# R

#### Instructions

Take after a meal with 16 oz of fluid, twice a day, 160mg



Stuc Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS\_001\_0016432874 9:41 ••• ■• My Plan



Date August 10, 2021



#### 12.14 Notifications

9:41



# Want to turn on notification reminders?

We'll remind you to complete your daily log for your doctor as well as notify you about new messages or requests from your care team.





# 12.15 Settings



#### Date August 10, 2021



#### Date August 10, 2021



Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4 Date August 10, 2021

| No SIM <b>奈</b> | 10:08 AM |
|-----------------|----------|
| Back | Profile |
| Mobile Phone | Number |
| Mobile Priorie | Number |
| +1(123)-456 | -7890 |
| | Save |

#### **12.16** Trends



# Dec 06 - Dec 12







< Symptoms

6

Medications >

10

11

9

< Medications

2.0 L

11

#### **Date August 10, 2021**



#### Dec 06 - Dec 12





11

Dec 06 - Dec 12



Dec 06 - Dec 12



Feeling >

# 12.17 Study Ending



My plan

Trends

Messages

Settings





### **Study Ending**

This study ends on Thursday, November 19, 2020. The app will not be available to use after that date.

Thank you for being part of this study. Your participation will help others living with heart failure.

If you have any questions about the study or the app, contact PPD , the Clinical Research Coordinator.







# **Study Ended**

The study you have been participating in is now closed. Thank you for your participation, and generous contribution to healthcare.

If you have any questions please contact PPD , the Clinical Research Coordinator. We will inform you once this platform is offered to all patients, at which point you will be able to continue your use.



#### 13. APPENDIX F. CLINICAL CASE REPORT FORM

# **Clinical Case Report Form**

| Screening ID | |
|---|---|
| Participant ID | |
| BI linked ID | |
| Date of Enrollment | |
| Confirmation of Eligibility Into the Stud | ly |
| Patient is $\geq 18$ years of age at the time of e<br>Yes<br>No | enrollment? |
| Patient diagnosed with asthma?<br>Yes<br>No | |
| | rnet access with the following requirements: iOS evices iPhone 8 or newer) or Android (Operating |
| Patient is able to understand and speak Enpatient app? Yes No | glish sufficiently to be able to use the AMAZE <sup>TM</sup> |
| Patient provided consent to participate?<br>Yes | |

Does the patient have a cognitive impairment, hearing difficulty, visual impairment, acute psychopathology, medical condition, or insufficient knowledge of the English language that, in the opinion of the investigator or interviewer, would interfere with his or her ability to provide electronic consent and/or participate/complete the questionnaire?

Yes

No

Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4 Date August 10, 2021 No (If yes - patient CANNOT be enrolled into the study) Investigator/Coordinator Full Name Dawei Jiang Remona Kanyat Dalton Lancaster Peter Moschovis Jehan Alladina Investigator/Coordinator Signature: Date: Did the patient download the AMAZE DMP App? \_\_\_\_\_ yes, \_\_\_\_\_ no IF YES, please record the BrightInsight ID Number: (Add a comment if BI ID has not been provided yet.) **Patient Characteristics** Age (years): \_\_\_ | Height: ft in; Weight: lb Sex:  $\square$  Male  $\square$  Female **ASTHMA DIAGNOSIS** Age when first diagnosed with asthma: (Years (if unknown, please mark the box below)) ☐ Unknown Duration patient seen by a health care provider for asthma: years months Duration patient seen by a healthcare provider at MGH for asthma: years months Smoking status (tobacco products, electronic cigarettes, vaping, marijuana) Smoking Status □ Never smoked □ Previously Smoker □ Current Smoker Previously smoked □ Cigarettes □ Vaping □ Marijuana Number of years smoked Average cigarette packs/vaping or marijuana times per day: Choose an option to Record "Time Since Last Smoke" ☐ Weeks ☐ Months ☐ Years Time since last smoked: Weeks \_\_\_\_\_ (Weeks) Months \_\_\_\_\_ (Months) Years \_\_\_\_ (Years) Currently smoking □ Cigarettes □ Vaping □ Marijuana

Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4 Date August 10, 2021

| Number of years smoked | (Years) |
|---|---|
| Average cigarette packs/vaping or marijuana times per day: | |
| Date last smoked:(Date) | |
| Time last smoked: (Time) | |
| Was spirometry lung function testing perfor | med on this nations in the last 12 months? |
| Yes □ No | med on this patient in the last 12 months: |
| Date of the most recent Spirometry test | |
| FEV1: Liters (Liters) | |
| FEV1: % Predicted ( | % Predicted) |
| FEV1: % Predicted (Liters) | |
| FVC: % Predicted (% | % Predicted) |
| FEV1:FVC: | |
| FEV1:FVC: FEV1/FVC: % Predicted | (% Predicted) |
| Was a test for eosinophil blood count perfor | med on this patient in the last 12 months? |
| ☐ Yes ☐ No | _ |
| Date of highest Absolute Eosinophil Count | Test(Absolute Eosinophil Count) |
| Absolute Eosinophil Count (Highest) | (Absolute Eosinophil Count) |
| How would you rate this patient's asthma se | everity? |
| ☐ Intermittent | |
| ☐ Mild persistent | |
| ☐ Moderate persistent | |
| Severe persistent | |
| At the last visit, do you think patient was: | NO ER visit and NO steroid prescriptions in the |
| past 12 months) | TWO ER VISIT and INO Steroid prescriptions in the |
| , | , and 1 ER visit or 1 steroid prescription in the past |
| 12 months) | , and I Lik visit of I sterota prescription in the past |
| ☐ Very poorly controlled (1+ hospitalization | n_and/or 2+ FR_visits_and/or 2+ steroid |
| prescriptions in the past 12 months) | ii, and of 2.1 Dit visits, and of 2.1 storoid |
| MAINTENANCE PHARMACOLOGIC THERA | PV |
| | currently prescribed and taking. Please check all that apply. |
| ICS | LAMA |
| ☐ QVAR HFA/Redihaler (beclomethasone | ☐ Incruse Ellipta (Umeclidinium) |
| dipropionate) | ☐ Spiriva Respimat/Handihaler (tiotropium bromide) |
| ☐ Beclovent HFA (beclomethasone | ☐ Tudorza/Aclidinium (aclidinium bromide) |
| dipropionate) | Triple Therapy (fixed dose combination) |
| ☐ Vanceril HFA) (beclomethasone dipropionate) | ☐ Trelegy Ellipta (fluticasone/umeclidinium/vilanterol) |
| ☐ Pulmicort Flexhaler/Respules (budesonide) | LTRA |
| Aerospan (flunisolide) | |
| ☐ Flunisolide ☐ Singulair (Montelukast) ☐ Flunisolide ☐ Accolate (Zafirlukast) | |
| ☐ Flovent HFA/Disc (fluticasone propionate) | ☐ Zyflo (Zileuton) |

| MAINTENANCE PHARMACOLOGIC THERAPY | |
|---|---|
| Please only include current medication the patient is currently prescribed and taking. Please check all that apply. | |
| ☐ Azmanex Twisthaler/HFA (mometasone | Theophylline Preparations |
| furoate) | ☐ Theo-24 (Theophylline) |
| ☐ Arnuity Ellipta (fluticasone furoate inhalation | ☐ Elixophylline (Theophylline) |
| powder)) | ☐ Theochron (Theophylline) |
| ☐ Triamcinolbone Acetonide | Chronic Add-on Therapy (Macrolides) |
| □ Alvesco | ☐ Zithromax (Azithromycin ) |
| ICS/LABA | ☐ Biaxin (Clarithromycin) |
| ☐ Advair Diskus/HFA (fluticasone propionate and | ☐ Erythromycin (Erythrocin) |
| salmeterol) ☐ Wixela Inhub (fluticasone propionate and | Biologics |
| salmeterol) | ☐ Cinqair (reslizumab) |
| ☐ Airduo Respiclick (fluticasone propionate and | ☐ Dupixent (dupilumab) |
| salmeterol) | ☐ Fasenra (benralizumab) |
| ☐ Breo Ellipta (fluticasone furoate and vilanterol) ☐ Dulera HFA (mometasone furoate and | ☐ Nucala (mepolizumab) |
| formoterol fumarate dihydrate) | ☐ Xolair (omalizumab) |
| ☐ Symbicort (budesonide/formoterol fumarate | |
| dihydrate) □ Budesonide/formoterol | |
| LABA (Single inhaled medicine, <i>not</i> in a fixed dose combination with an ICS or ICS/LAMA) | |
| dose comonation with an 105 of 105/2/1911) | |
| ☐ Serevent (Salmeterol xinafoate) | |
| ☐ Foradil (formoterol fumarate) | |
| ☐ Arcapta (Indacaterol) | |
| ☐ Brovana (arformoterol tartrate) | |
| ☐ Indacaterol | |
| ☐ Arformoterol ☐ Striverdi (Oldaterol) | |
| SABA/Rescue Inhaler Use | |
| ☐ Daily Use (SABA) | |
| ☐ SABA alone | |
| □ SABA+ICS | |
| □ LABA+ICS | |
| □ Nebulizer | |
| Nebulizer – Please Specify | |
| recounted – Flease specify | |
| ☐ Other – Please Specify | |
| Which of the following did you do to the patient's m | edication after their LAST visit? (Check all that apply) |
| ☐ Step-down of controller medicines | ( 11 7) |
| ☐ No change of controller medicines | |
| ☐ Step-up of controller medicines | |
| ☐ Prescribe a course of systemic corticosteroids | |

Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4 Date August 10, 2021

| MAINTENANCE PHARMACOLOGIC THERAPY |
|---|
| Please only include current medication the patient is currently prescribed and taking. Please check all that app |
| □ Other: |
| Investigator Final Confirmation |
| Investigator/Coordinator Signature: |
| Date: |
| 14. APPENDIX G. PATIENT DEMOGRAPHIC QUESTIONNAIRE |
| Demographic Questionnaire (AMAZE <sup>TM</sup> App) |
| Dear Research Participant, |
| Thank you for taking part of the AMAZE <sup>TM</sup> Asthma Research Study at Massachusetts General Hospital (MGH). |
| As part of the study procedure, please complete the survey below. |
| If you have any questions, please contact the Study Team at CCI. |
| Thank you! |
| What is your age? (years) |
| What is your biological sex? |
| ☐ Male ☐ Female |
| What is your ethnic background? |
| <ul> <li>☐ Hispanic or Latino</li> <li>☐ Not Hispanic or Latino</li> <li>☐ Prefer not to say</li> </ul> |
| What is your racial background? |
| Study Protocol Form |

| Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4 Date August 10, 2021 White Black or African American Asian Native Hawaiian or other Pacific Islander American Indian or Alaska Native Other (specify): |
|---|
| □ Prefer not to say |
| What is your current living/domestic situation? |
| <ul> <li>☐ Living alone</li> <li>☐ Living with a spouse, partner, family, or friends</li> <li>☐ Other (specify):</li> </ul> |
| How would you describe your employment status? |
| <ul> <li>□ Employed, full-time</li> <li>□ Employed, part-time</li> <li>□ Homemaker</li> <li>□ Student</li> <li>□ Unemployed</li> <li>□ Retired</li> <li>□ Disabled</li> <li>□ Other (specify):</li> </ul> |
| What is the highest level of education you have completed? Less than high school Secondary/high school Associate degree, technical or trade school College/university degree Postgraduate school Other (specify): |
| What is your household's total income from all sources over the past 12 months? |
| ☐ Less than \$15,000 ☐ \$15,000 to \$29,999 ☐ \$30,000 to \$44,999 ☐ \$45,000 to \$59,999 ☐ \$60,000 to \$74,999 ☐ \$75,000 to \$99,999 ☐ \$100,000 or more ☐ Prefer not to answer |
| Age when you were first diagnosed with asthma? (year-old) |
| Study Protocol Form<br>Version 7.4 |

St Form Doc ID: AZDoc0059948
Parent Doc ID: SOP LDMS\_001\_0016432892 Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4 Date August 10, 2021

| How many years (and months) seen by a health care provider for asthma with asthma |
|---|
| (years (and months)) |
| How many years (and months) seen by a MGH provider for asthma with asthma (years (and months)) |
| Do you currently smoke? |
| ☐ Yes, smoker ☐ Not currently, but previous smoker ☐ No, never smoked |
| Do you currently vape? ☐ Yes, vaper |
| ☐ Not currently, but previous vaper ☐ No, never vaped |
| Do you have any of the following health conditions? (Check all that apply) |
| <ul> <li>□ No other health conditions</li> <li>□ Allergy diagnosed by blood or skin testing</li> <li>□ Allergic rhinitis (nasal allergies, "hay fever")</li> <li>□ Heart disease (history of heart attack, heart failure or heart valve problems)</li> <li>□ Anxiety</li> <li>□ Anaphylaxis (severe allergic reaction to a food, bee sting, allergy shot, medication or other</li> <li>□ Arthritis</li> <li>□ Aspirin sensitivity (aspirin causes hives, swelling or breathing problems)</li> <li>□ Atopic dermatitis/Eczema</li> </ul> |
| ☐ Chronic bronchitis ☐ Chronic Obstructive Pulmonary Disease (COPD) ☐ Chronic sinusitis ☐ Depression ☐ Diabetes ☐ Emphysema ☐ GERD (heartburn/reflux) |
| ☐ Hypertension (high blood pressure) ☐ Nasal Polyps ☐ Sleep Apnea tudy Protocol Form |
| Yersion 7.4 |

| tudy Protocol |
|---|
| tudy Code D2287R00166 [EVA-28838] |
| Version 7.4 Date August 10, 2021 |
| □ Stroke |
| ☐ Other (specify): |
| □ Don't know |
| Do you currently have health insurance? |
| □ Yes |
| □ No |
| ☐ Prefer not to answer |
| Programmer note: If answered "yes"] What type of health insurance coverage do you have? Check all that apply) |
| ☐ Third-party payer (for example, United Healthcare, Blue Cross/Blue Shield, Aetna.) |
| ☐ Managed care organization |
| ☐ Tricare (military health insurance) |
| ☐ Medicare |
| ☐ Medicaid (MassHealth) |
| □ Self-pay |
| □ Unsure |
| ☐ Other (please specify): |

# 15. APPENDIX H. PATIENT VISIT EXPERIENCE SURVEY

| Visit Experience Survey (A | MAZETM | (App) | | | | |
|---|---|---|---|---|---|---|
| Dear Research Participant, | | | | | | |
| Thank you for taking part of the A Hospital (MGH). | AMAZE <sup>TM</sup> A | Asthma Res | search St | udy at Mas | ssachusetts | General |
| As part of the study procedure, pl | ease comple | ete the surv | ey below | | | |
| If you have any questions, please | contact the | Study Team | n at <mark>CCI</mark> | | | |
| Thank you! | | | | | | |
| You've been using the AMAZE <sup>TM</sup><br>on asthma. Please answer the fol<br>App may have affected your clinic | lowing ques | tions, keepi | ng in mi | | | |
| Your responses are strictly confi | dential and | will not aff | ect your | clinical co | are in any w | vay. |
| 1) Was the visit initiated by (chec | ck one): | | | | | |
| ☐ Patient | | | | | | |
| ☐ Healthcare Provider | | | | | | |
| | | Strongly<br>Agree | Agree | Neutral | Disagree | Strongly<br>Disagree |
| 2) The AMAZE <sup>TM</sup> App<br>helped me discuss my asthma<br>with my healthcare<br>provider(s) during my most<br>recent visit | □ Not applicable | | | | | |
| 3) I received information about my asthma that helped me better understand my | □ Not applicable | | | | | |

 $\square$  Not

applicable

 $\square$  Not

applicable

condition during my most

4) I received information

about my asthma medications

during my most recent visit

5) I was given information

about additional care that I

recent visit

| need for my asthma during my most recent visit | |
|---|---|
| 6) I was included in making decisions about my asthma treatment during my most recent visit | □ Not applicable |
| 7) The AMAZE <sup>TM</sup> <i>App</i> helped the appointment with my doctor go more smoothly. | □ Not applicable |
| 8) The time spent with my healthcare provider(s) discussing my asthma during my most recent visit was better compared to my last visit. | □ Not applicable |
| 9) I found it was easier to schedule an appointment with my doctor using the AMAZE <sup>TM</sup> App | □ Not applicable |
| 10) The visit helped avoid an ER or Urgent Care center visit or hospitalization | □ Not applicable |

#### 16. APPENDIX I. POST-STUDY SURVEY (FOR HCPS)

# Post-Study Survey (AMAZE<sup>TM</sup> App - Clinical Staff Research Participant)

Dear Clinical Staff Research Participant,

Parent Doc ID: SOP LDMS\_001\_0016432897

Thank you for taking part of the AMAZE<sup>TM</sup> Asthma Research Study at Massachusetts General Hospital (MGH).

As part of the study procedure, please complete the survey below.

If you have any questions, please contact the Study Team at CCl Thank you!

The purpose of this questionnaire is to obtain your feedback on the implementation of AMAZE<sup>TM</sup>. This questionnaire should take approximately 10 minutes to complete. As an employee of MGH, your participation is completely voluntary and will not impact your job in a positive or negative manner. All information collected from you will be kept without any personal information. You will be identified in the research records by a code name or number. By completing this questionnaire, you are agreeing to participate in this study.

| | How would you rate the overall ease of implementing AMAZE $^{\text{\tiny TM}}$ on a platform into your clinical practice? |
|---|---|
| | <ul> <li>□ Very easy</li> <li>□ Somewhat easy</li> <li>□ Not easy or difficult</li> <li>□ Difficult</li> <li>□ Very Difficult</li> </ul> |
| | Did the AMAZE <sup>™</sup> help you manage your patients? |
| | □ Not at all □ Slightly □ Somewhat □ Moderately □ Very well |
| | Regardless of intermittent or persistent, on average, what percentage of your asthma patients would you classify as: |
| Vers | % Mild asthma% Moderate asthma% Severe asthma = 100% y Protocol Form iion 7.4 n Doc ID: AZDoc0059948 |

Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4 Date August 10, 2021

| On average, what percentage of your patients would you classify as: |
|---|
| Well-controlled % Not well-controlled % Very poorly controlled = 100% |
| On average, what percentage of your asthma patients do you feel are at (1) low, (2) medium, and (3) high risk for adverse outcomes from their asthma? Please fill out below. % Low risk % Medium risk % High risk |
| = 100% |
| Did AMAZE <sup>TM</sup> help you identify patients who were at risk for adverse health outcome (e.g., hospitalizations, exacerbations, medication side effects) from their asthma that you would have otherwise missed? |
| □ Yes □ No |
| What did you find most useful about the AMAZE <sup>TM</sup> platform? Check all that apply |
| <ul> <li>□ Ability to asthma triggers</li> <li>□ Ability to track reliever medication use</li> <li>□ Ability track ER visits/ hospitalizations</li> <li>□ Ability to track air flow measurements</li> <li>□ Patient-HCP messaging feature</li> <li>□ Ability to assign another healthcare provider to a patient</li> <li>□ Integration of AMAZE<sup>TM</sup> platform with electronic health records</li> <li>□ Ability to track level of impairment through ACT<sup>TM</sup> scores</li> <li>□ Ability to receive alerts (flags) based on patient responses in the app</li> <li>□ Other:</li> </ul> |
| What did you find <u>least</u> useful or cumbersome about AMAZE <sup>TM</sup> platform? <i>Check all that apply</i> |
| ☐ Ability to track symptoms |
| y Protocol Form |

Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4

| Date | August | 10, | 2021 |
|------|--------|-----|------|
|------|--------|-----|------|

| ☐ Ability to track level of impa | talizations surements are lthcare provider to a patient atform with electronic health records irment through ACT <sup>TM</sup> scores s) based on patient responses in the app |
|---|---|
| How frequently would you want<br>patients?<br>Symptoms<br>Asthma triggers<br>Rescue medication use<br>Maintenance medication use<br>Steroid medication use<br>ER / Urgent Care visits<br>Peak flow / FEV1 | to track the following for appropriate management of Daily Weekly Monthly Other Daily Meekly Monthly Other Daily Meekly Monthly Other |
| ☐ Increased recognition of patien ☐ Increased recognition of conce ☐ Improved recognition of patien ☐ Improved recognition of patients. | t with their treatment, risk, or control with their treatment |
| While using AMAZE <sup>TM</sup> disease treatment? | management platform (DMP), how often did you change |
| ☐ Step up (for exam | |

Study Protocol Study Code D2287R00166 [EVA-28838] Version 7.4 Date August 10, 2021

| What features of AMAZE <sup>TM</sup> do you think could be imp | roved? |
|---|---|
| | _ |
| | _ |
| | _ |
| What barriers did you encounter in implementing AMA | ZE <sup>TM</sup> into your clinical practice |
| | _ |
| | _ |
| Do you have any other comments or suggestion? | |
| Do you have any owner comments of suggestion. | |
| | _ |
| | _ |

# 17. APPENDIX J. PATIENT SATISFACTION QUESTIONNAIRE-18 (PSQ-18)

# Participant Satisfaction Questionnaire-18 (PSQ-18)

Dear Research Participant,

Thank you for taking part of the AMAZE<sup>TM</sup> Asthma Research Study at Massachusetts General Hospital (MGH).

As part of the study procedure, please complete the survey below.

If you have any questions, please contact the Study Team at CCI Thank you!

In the table below are some things people say about medical care. Please read each one carefully, keeping in mind the medical care you are receiving now. (If you have not received care recently, think about what you would expect if you needed care today.) We are interested in your feelings, good and bad, about the medical care you have received.

# SHORT-FORM PATIENT SATISFACTION QUESTIONNAIRE (PSQ-18)

These next questions are about how you feel about the medical care you receive.

On the following pages are some things people say about medical care. Please read each one carefully, keeping in mind the medical care you are receiving now. (If you have not received care recently, think about what you would <u>expect</u> if you needed care today.) We are interested in your feelings, good and bad, about the medical care you have received.

How strongly do you AGREE or DISAGREE with each of the following statements?

(Circle One Number on Each Line)

| | | Strongly<br><u>Agree</u> | Agree | Uncertain | Disagree | Strongly<br>Disagree |
|---|---|---|---|---|---|---|
| 1. | Doctors are good about explaining the reason for medical tests | 1 | 2 | 3 | 4 | 5 |
| 2. | I think my doctor's office has<br>everything needed to provide<br>complete medical care | 1 | 2 | 3 | 4 | 5 |
| 3. | The medical care I have been receiving is just about perfect | 1 | 2 | 3 | 4 | 5 |
| 4. | Sometimes doctors make me wonder if their diagnosis is correct | 1 | 2 | 3 | 4 | 5 |
| 5. | I feel confident that I can get the medical care I need without being set back financially | 1 | 2 | 3 | 4 | 5 |
| 6. | When I go for medical care, they are careful to check everything when treating and examining me | 1 | 2 | 3 | 4 | 5 |
| 7. | I have to pay for more of my medical care than I can afford | 1 | 2 | 3 | 4 | 5 |
| 8. | I have easy access to the medical specialists I need | 1 | 2 | 3 | 4 | 5 |

# How strongly do you AGREE or DISAGREE with each of the following statements?

(Circle One Number on Each Line)

| | | Strongly<br>Agree | Agree | Uncertain | Disagree | Strongly<br><u>Disagree</u> |
|---|---|---|---|---|---|---|
| 9. | Where I get medical care, people have to wait too long for emergency treatment | 1 | 2 | 3 | 4 | 5 |
| 10. | Doctors act too businesslike and impersonal toward me | 1 | 2 | 3 | 4 | 5 |
| 11. | My doctors treat me in a very friendly and courteous manner | 1 | 2 | 3 | 4 | 5 |
| 12. | Those who provide my medical care sometimes hurry too much when they treat me | 1 | 2 | 3 | 4 | 5 |
| 13. | Doctors sometimes ignore what I tell them | 1 | 2 | 3 | 4 | 5 |
| 14. | I have some doubts about the ability of the doctors who treat me | 1 | 2 | 3 | 4 | 5 |
| 15. | Doctors usually spend plenty of time with me | 1 | 2 | 3 | 4 | 5 |
| 16. | I find it hard to get an appointment for medical care right away | 1 | 2 | 3 | 4 | 5 |
| 17. | I am dissatisfied with some things about the medical care I receive | 1 | 2 | 3 | 4 | 5 |
| 18. | I am able to get medical care whenever I need it | 1 | 2 | 3 | 4 | 5 |

# 18. APPENDIX K. SIX-MONTH CHART REVIEW CASE REPORT FORM



Date August 10, 2021

New Medication/ Continued, Same Dose/ Continued, Increased Dose/ Continued, Decrease Dose/ Discontinued/ Not Applicable

ICS - Aerospan (flunisolide)

ICS - Alvesco (ciclesonide)

ICS - Arnuity Ellipta (fluticasone

furoate inhalation powder)

ICS - Asmanex Twisthaler/HFA

(mometasone furoate)

ICS - Beclovent HFA

(beclomethasone dipropionate)

ICS - Flovent HFA/Disc

(fluticasone propionate)

ICS - Flunisolide

ICS - Pulmicort

Flexhaler/Respules (budesonide)

ICS - QVAR HFA/Redihaler

(beclomethasone dipropionate)

ICS - Triamcinolone Acetonide

ICS - Vanceril HFA

(beclomethasone dipropionate)

ICS/LABA - Advair Diskus/HFA

(fluticasone propionate and

salmeterol)

ICS/LABA - Airduo Respiclick

(fluticasone propionate and

salmeterol)

ICS/LABA - Breo Ellipta

(fluticasone furoate and

vilanterol)

ICS/LABA -

IBCuSd/eLAsoBnAi d-e D/fuolremrao tHeFrAol

(mometasone furoate and

formoterol fumarate dihydrate)

ICS/LABA - Symbicort

(budesonide/formoterol

fumarate dihydrate)

ICS/LABA - Wixela Inhub

(fluticasone propionate and

salmeterol)

LABA - Arcapta (Indacaterol)

LABA - Arformoterol

LABA - Brovana (arformoterol

tartrate)

LABA - Foradil (formoterol

fumarate)

LABA - Indacaterol

LABA - Serevent (Salmeterol

xinafoate)

LABA - Striverdi (Oldaterol)

Study Protocol Form

Version 7.4

Form Doc ID: AZDoc0059948

Parent Doc ID: SOP LDMS 001 00164328105

LAMA - Incruse Ellipta

(Umeclidinium)

LAMA - Spiriva

Respimat/Handihaler (tiotropium

bromide)

LAMA - Tudorza/Aclidinium

(aclidinium bromide)

Triple Therapy (fixed dose

combination) - Trelegy Ellipta

(fluticasone furoate,

umeclidinium, vilanterol)

LTRA - Accolate (Zafirlukast)

LTRA - Singulair (montelukast

sodium)

LTRA - Zyflo (zileuton)

Theophylline Preparations -

Elixophylline (Theophylline)

Theophylline Preparations -

Theo-24 (Theophylline)

Theophylline Preparations -

Theochron (Theophylline)

Chronic Add-on Therapy

(Macrolides) - Zithromax

(Azithromycin)

Chronic Add-on Therapy

(Macrolides) - Biaxin

(Clarithromycin)

Chronic Add-on Therapy

(Macrolides) - Erythromycin

(Erythrocin)

Biologics - Cinqair (reslizumab)

Biologics - Dupixent (dupilumab)

Biologics - Fasenra

(benralizumab)

Biologics - Nucala

(Bmioelopgoilcizsu -m Xaobla)ir (omalizumab)

Rescue Inhaler Use - Daily Use

(SABA)

Rescue Inhaler Use - SABA alone

Rescue Inhaler Use - SABA+ICS

Rescue Inhaler Use - LABA+ICS

Rescue Inhaler Use - Nebulizer

Rescue Inhaler Use - SAMA

Other - Please specify

Name of Nebulizer

# **ASTHMA EXACERBATION HISTORY**

| steroid<br>and/or<br>Impor<br>count | thma exacerbation is defined by a change in asthma control requiring a course of oral ds (i.e., at least 3 days with at least 10 days between each burst) and/or steroid injection r a hospitalization or emergency department visit for an asthma exacerbation. retantly, record only the highest utilization for each exacerbation, do not double exacerbation episodes. If an OCS course was due to a hospitalization, do not record CS course but as the hospitalization |
|---|---|
| 4. | Number of times since enrollment asthma symptoms required an emergency department or urgent care visit (but not an overnight stay in the hospital): |
| | ER/urgent care visits (with no overnight hospital stay) |
| 5. | Number of times since enrollment that there was a worsening in asthma symptoms that required a hospital stay for greater than 24 hours: times admitted to hospital |
| 6. | Number of unplanned ambulatory clinic visits due to exacerbation in since enrollment: unplanned visits |
| 7. | How many courses of oral corticosteroids (OCS) was the patient prescribed over the since enrollment for asthma exacerbations unrelated to emergency department, urgent care or, unplanned ambulatory clinic visits or hospitalizations? |
| Investi | gator Final Confirmation |
| Investig | gator/Coordinator Full Name |
| Dalton<br>Peter M | Jiang<br>a Kanyat<br>Lancaster<br>Ioschovis<br>Alladina |
| | gator/Coordinator Signature: |
| Date: | |

# 20. APPENDIX L. MGH WORKFLOW FOR IMPLEMENTATION OF DMP IN CLINICAL PRACTICE

#### Screening:

 $\sim$ 33 young adults (18–35 yr) and up to 17 adults (>=36 yr).

#### **Inclusion Criteria:**

- >=18 yr with Dx of asthma (with or without COPD).
- Own smartphone with compatible OS.
- Able to sufficiently use the AMAZE™ patient App.
- Consenting to participate in the study procedures.

#### **Exclusion Criteria:**

- No current diagnosis of asthma.
- Cognitive impairment, hearing difficulty, insufficient knowledge of English, or any medical condition interfering with study participation.

#### **Enrollment:**

- eConsent via REDCap.
- Download AMAZE™ App, set up account, provided with a unique identifier.

#### **Baseline Visit:**

- Patient to complete sociodemographic form.
- Staff will complete a clinical CRF in REDCap.

#### Patient to complete:

- Daily log
- ACT™ (every four weeks)
- Patient User Experience Survey (months 1, 3, and 6 via email)
- Patient Visit Experience Survey (after each in-person or telehealth clinic visit )
- System Usability Scale (months 1 and 6)
- Patient Satisfaction Questionnaire-18
- 12 patients for longitudinal interviews at months 1, 3, and 6;
- 5 patients for one cross-sectional interview at months 2, 4, or 5.
# MGH staff to complete:

- Clinical Case Report Form (initial visit)
- Chart Review Case Report Form (month 6)
- System Usability Scale (months 1 and 6)
- Follow-up Process Interviews (n=4, months 1, 3, and 6)
- Post-study Survey

## Study monitoring:

- Nurse to monitor the patient dashboard twice a day
- Physician to review the dashboard during every clinical visit

#### **Outcomes:**

Primary Outcome: Feasibility, usability, perceived value, and potential benefits of the AMAZE™ implemented in clinical practice.

Process Outcomes: Evaluating the impact of AMAZE™ on clinical practice, including duration of patient visits and services, as well as responses to survey items on changes to timing of scheduling visits, communication during the visit, and satisfaction with medical care received.

Exploratory Clinical Outcomes: evaluate how AMAZE impacts key clinical outcomes including exacerbations, HCRU, change in therapy, and exposure to COVID-19

# 21. APPENDIX M. PATIENT USER EXPERIENCE SURVEY

# User Experience Survey (AMAZE<sup>TM</sup> App)

| Dear Research Participant, |
|---|
| Thank you for taking part of the AMAZE <sup>TM</sup> Asthma Research Study at Massachusetts General Hospital (MGH). |
| As part of the study procedure, please complete the survey below. |
| If you have any questions, please contact the Study Team at CC. |
| Thank you! |
| In general, how would you describe your asthma in terms of severity? A. Mild B. Moderate C. Severe D. Other (Please specify): |
| Approximately, how many asthma flare-ups (also called exacerbations) did you have in the last 30 days? # of flare-ups |
| Who is your primary asthma doctor at Massachusetts General Hospital (MGH)? PPD |

| Study Protocol |
|------------------------------------|
| Study Code D2287R00166 [EVA-28838] |
| Version 7.4 |
| Date August 10, 2021 |

Overall, how satisfied are you with your asthma care at MGH?

Very Unsatisfied

Unsatisfied

Neutral

Satisfied

Very Satisfied

Indicate your level of agreement with the following statement:

I have control over my asthma.

Strongly Agree

Agree

Neither

Disagree

Strongly disagree

I understand my asthma.

Strongly agree

Agree

Neither agree nor disagree

Disagree

Strongly disagree

Since the start of the study, use of the AMAZE<sup>TM</sup> app helped me avoid ER or Urgent Care center visit(s) or hospitalization(s).

- A. Strongly agree
- B. Agree
- C. Neither agree nor disagree
- D. Disagree
- E. Strongly disagree
- F. Not applicable I did not use the app

Please **rate** the following features using a 5-point rating with 5 being the best possible score. If you do not use a given feature, you do not have to rate it.

1 (lowest score)
2
3
4
5 (highest score)
Did not use the feature
Study Protocol Form
Version 7.4
Form Doc ID: AZDoc0059948

Parent Doc ID: SOP LDMS\_001\_00164328111

Daily log (where you track symptoms, etc.)

Messaging with MGH

Asthma education (articles, videos)

Air quality

My Plan (list of meds & reminders)

Trends (daily log summaries / graphs)

Appointments (viewing and scheduling)

Care Team Request (Asthma Control Test<sup>TM</sup> - monthly 5-question survey)

How frequently do you want to track the following for your doctor:

| Symptoms | Daily | Weekly | Monthly | Other (Please Specify) |
|---|---|---|---|---|
| Asthma triggers | Daily | Weekly | Monthly | Other (Please Specify) |
| Rescue medication use | Daily | Weekly | Monthly | Other (Please Specify) |
| Maintenance medication use | e Dai | ly Week | dy Month | ly Other (Please Specify) |
| Steroid medication use | Daily | Weekly | Monthly | Other (Please Specify) |
| ER / Urgent Care visits | Daily | Weekly | Monthly | Other (Please Specify) |
| Peak flow / FEV1 | Daily | Weekly | Monthly | Other (Please Specify) |

What concerns if any do you have about the AMAZE<sup>TM</sup> app? [Select all that apply]

Data / privacy concerns.

I do not find the app helpful.

I forget to use it.

There are things missing that I want in the app.

It is not fun to use.

It is not easy to use.

Other:

[radio button] I do not have any concerns.

Overall, how satisfied are you with the AMAZE<sup>TM</sup> App?

Very Unsatisfied

Unsatisfied

Neutral

Satisfied

Very Satisfied

Why do you feel that way about the AMAZE<sup>TM</sup> App?

Study Protocol Form Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS 001 00164328112

How likely are you to recommend the AMAZE<sup>TM</sup> App to another patient at MGH who has asthma?

Very Unlikely

Unlikely

Undecided

Likely

Very Likely

Please share any additional feedback you have about the app (suggested topics below):

- What you like vs do not like about the app
- What works well vs what does not
- Any issues / bugs you have found in the app
- Anything else you think we should know about the app

# 22. APPENDIX N.1 SYSTEM USABILITY SCALE (SUS) ADMINISTERED AT MONTHS 1 AND 6: Patients

System Usability Scale Survey (AMAZE<sup>TM</sup> App)

Dear Research Participant,

Thank you for taking part of the AMAZE<sup>TM</sup> Asthma Research Study at Massachusetts General Hospital (MGH).

As part of the study procedure, please complete the survey below.

| Francisco Franci |
|---|
| If you have any questions, please contact the Study Team at CCI |
| Thank you! |
| For each of the following statements, mark one box that best describes your reactions to the AMAZE <sup>TM</sup> Application (App). |

**Strongly** Neutral Disagree Strongly Agree Agree Disagree I think that I would like to use this app frequently. I found the app unnecessarily complex. I thought the app was easy to use. I think that I would need the support of a technical person to be able to use this app. I found the various functions in this app were well integrated. I thought there was too much П П П inconsistency in this app. I would imagine that most people would П learn to use this app very quickly. I found the app very cumbersome to use. I felt very confident using the app. I needed to learn a lot of things before I could get going with this app.

# 23. APPENDIX N.2 SYSTEM USABILITY SCALE (SUS) ADMINISTERED AT MONTHS 1 AND 6: MGH Staff

System Usability Scale Survey (AMAZE<sup>TM</sup> App – Clinical Staff Research Participant)

Dear Clinical Staff Research Participant,

Thank you for taking part of the AMAZE<sup>TM</sup> Asthma Research Study at Massachusetts General Hospital (MGH).

As part of the study procedure, please complete the survey below.

If you have any questions, please contact the Study Team at CCI Thank you!

For each of the following statements, mark one box that best describes your reactions to the AMAZE<sup>TM</sup> clinician dashboard.

| | Strongly<br>Agree | Agree | Neutral | Disagree | Strongly<br>Disagree |
|---|---|---|---|---|---|
| I think that I would like to use this dashboard frequently. | | | | | |
| I found the dashboard unnecessarily complex. | | | | | |
| I thought the dashboard was easy to use. | | | | | |
| I think that I would need the support of a technical person to be able to use this dashboard. | | | | | |
| I found the various functions in this dashboard were well integrated. | | | | | |
| I thought there was too much inconsistency in this dashboard. | | | | | |
| I would imagine that most people would learn to use this dashboard very quickly. | | | | | |
| I found the dashboard very cumbersome to use. | | | | | |
| I felt very confident using the dashboard. | | | | | |
| I needed to learn a lot of things before I could get going with this dashboard. | | | | | |

# 24. APPENDIX O. FOLLOW-UP SEMI-STRUCTURED INTERVIEW GUIDES

## Longitudinal Follow-up Interview Guide [For months One, Three, and Six]

Hello, my name is [interviewer name] and I am working with [MGH] and AstraZeneca to see how well the new asthma app is working for you. You previously consented to participate in this study regarding the asthma app and you have been randomly selected to participate in up to three interviews periodically through the duration of the study (roughly 1, 3, and 6 months after you enrolled in the study). During each interview, we will ask for your feedback on the [MGH] asthma app that you have been using, including ease of use, suggestions for changes. There are no right or wrong answers; we'd like to hear your personal experience with the app.

I would like to have your permission to audio record this session. The recording will be used to help us improve the app and write a report about the things we talked about here today. The audio will be transcribed by a third-party vendor, TransPerfect, but any identifying information you say during the interview will be removed from the transcript. It will be kept confidential and your name will not be linked with your responses. If an adverse event (side effect) for an AstraZeneca product were to come up during the course of this interview, I am required to report that.

Begin Recorder: This is participant ID [Insert number here] for [month one/three/six] longitudinal follow-up interview of study EVA-28838. Do I have your permission to record this session? I want to confirm that you still consent to participate in the interview.

Thank you for completing the asthma app so far.

#### Introduction

First, we'll be going over a brief introduction to your experience with medical apps and your smartphone.

- 1. How long have you have been using the asthma app?
- 2. When you initially started the study, you had an [iPhone or Android]. Just to confirm, do you still have that phone?
- 3. Do you use any medical health apps beside the asthma app?
  - a. [If needed]: If yes, what do you use and what do you use it for?

#### Asthma App – App Use and Experience

Now I'd like to ask you a few questions on your overall thoughts on the app and the notification/reminder system.

- 1. Overall, what do you think of the app?
  - a. In what ways is it easy to use?
  - b. In what ways is it hard to use?

- 2. [For month 1 interview only]: What did you think about the app when you were first contacted by [MGH]?
  - a. Walk me through the process of finding, downloading, and using the app.
  - b. Was there anything confusing or difficult for downloading the app and gaining access to the features?
- 3. Is there anything confusing about using the asthma app?
  - a. [If yes]: What is confusing?
- 4. Do you have any trouble accessing any of the features in the app?
  - a. [If yes]: Tell me more about that. What trouble do you have?
- 5. What notifications or reminders, if any, do you receive from the asthma app?
  - a. Do you find the reminders helpful?
    - i. Do you recall what time of day you set the reminders for? Why did you choose that time?
    - ii. [Probe as needed]: Do you recall what you received a reminder for (i.e., medications, daily log, air quality alerts)?
  - b. [If no]: Did you turn your notifications off? Would daily reminders have been helpful?
- 6. How often did you use the app? What time of day did you use it?
  - a. [*If less than once a day*]: Why did you use it less than once a day? Is there anything missing that would have made you more likely to use the app every day?
- 7. How, if at all, did you report issues/problems that you found in the app? (*Note to interviewer: there is an option for participants to report bugs/issues in the app.*)

### **Features of the App**

1. What features of the Asthma App (i.e., daily log, trends, messaging) do you use?

Now I'd like to go through each of the features with you. Feel free to open your app while we go through the sections. [Interviewer to wait for participant to open app if needed.]

- a. Interviewer for each of the features go through the following probes:
  - i. Do you use this feature in the app? If yes, how often do you use the app? If no, why do you not use this feature?
  - ii. How helpful is the feature? Would you continue to use this feature to help monitor your asthma?
  - iii. Is there anything confusing or unclear about this feature? What ideas do you have to make the feature better?
  - iv. [For daily log only]: Have you ever had to change any of your answers for the daily log? If so, did you have any problems making changes?
  - v. [For daily log only]: What did you think about the amount of time it took you to complete the daily log? Was it too long, too short, or enough time?

Study Protocol Form Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS 001 00164328117

| Feature | Use | Helpfulness | Suggestions |
|---------------|-----|-------------|-------------|
| Daily Log | | | |
| Air Quality | | | |
| Appointments | | | |
| ACT | | | |
| Education | | | |
| My Plan | | | |
| Trends | | | |
| Messaging | | | |
| Notifications | | | |

### **Text and Image Size**

- 4. Did you have any problems with the font size on any of the screens?
  - a. Would you change anything about the way the text or images appear on any of the screens?

### Using the App to Communicate with Doctor or During Visits

Now I'd like to discuss how you used the app to communicate with your doctor via the messaging feature or during a doctor's visit.

[Note to interviewer: the previous section probes on the messaging feature so use these probes if not fully addressed to this point.]

- 1. How do you typically communicate with your doctor outside of appointments?
- 2. Did you use the messaging feature to send communication to your doctor?
  - a. If yes, what things did you discuss while messaging your doctor?
    - i. Would you continue to use the messaging feature in the future? Why or why not?
    - ii. How often did you send messages to your doctor through the app?
    - iii. Which subject line did you typically use and why? [Note to interviewer: if needed explain that there is a forced choice for the subject line.]
  - b. If no, why did you not use the messaging feature?

- 3. We noticed you had a doctor's visit on [insert date]. Did you and your doctor discuss anything regarding the app during the visit?
  - a. If yes, what was discussed? Did you open the app during your visit and show any specific log or trends?
    - i. How did the app change the communication with your doctor during the visit compared to previous visits?
  - b. If no, do you think discussing the app or any feature of the app would have been helpful during your visit?

#### Long-Term Use

- 1. Would you consider using this app as a part of your long-term asthma care? Why or why not?
  - a. If no, what would improve your experience with completing this app every day?
- 2. What do you hope to gain from the app? What do you think your doctor will gain from you using the app?
- 3. Do you feel like using the app has helped you avoid ER or hospital visits? Why or why not?
- 4. Are you likely to recommend this app to a person living with asthma? Why or why not?
- 5. What other feedback would you like to give us on this app today?

Thank you! We are all done with the interview. Interviewer should confirm the participant still has a ClinCard and let them know the \$[insert payment] will be uploaded within 24 hours of the interview.

# Cross-Sectional Patient Discussion Guide: AMAZE<sup>TM</sup> Asthma App

- **Purpose.** Hi, my name is [\_\_\_\_] and I'm a researcher with AstraZeneca, a pharmaceutical company. We wanted to speak with you today to get your feedback on the AMAZE<sup>TM</sup> asthma app that you have been using. We want to know what you think of the app so we can continue making this app better for people like you.
- Anonymity / Confidentiality. The research is all confidential and anonymous and none of your data will be directly paired to you. To keep things confidential, please never say your full name or any other identifiable information like your phone number or address, etc. We'll stick to first names only.
- **Honest Feedback.** Feel free to provide your honest feedback about the app today. Don't be afraid to share negative feedback, if you have any. I didn't personally create this so it won't hurt my feelings.
- Adverse Events. I'm not here to sell or market you any drug, but, if you should mention you had an adverse reaction come up on an AstraZeneca drug, I am required for

compliance reasons to report any details of that event you experienced.

• Questions. Do you have any questions for me before we get started?

#### Patient Intro

- 1. Tell me a little about yourself what keeps you busy?
- 2. How long have you been living with asthma?
  - a. How would you characterize it: mild, moderate, severe?
- 3. What are some of the biggest challenges you face living with asthma?

## **Phone Type + Health Apps**

- 1. What type of phone do you have? I.e., Apple, Android?
- 2. How do you typically use your phone? What apps do you use the most?
- 3. Besides the asthma app, what kind of health apps/tools do you use or have you used in the past?
  - a. Examples: Think AppleHealth, Fit Bit, Clinician portal, Headspace, etc.
- 4. Do you use MyChart? If so, how?

# Experience with AMAZE<sup>TM</sup>

## **App Introduction**

- 1. How did you first learn about the asthma app?
  - a. What was your reaction when you heard about it?
  - b. Why do you think your clinician(s) wanted you to use the asthma app?
  - c. What made you decide to join the asthma study?

### **Onboarding**

- 2. Can you walk me through the process of finding and getting started with the app?
  - a. Who, if anyone, helped you get started with the app? i.e., caregiver, staff, doctor
  - b. How easy / difficult was it for you to find the app? How did you find it?
  - c. How easy / difficult was it for you to create an account?
  - d. What issues, if any, did you encounter with getting started with the app?
    - i. I.e., finding it, downloading it, creating an account, etc.
- 3. Is there anything that could have been done differently to make onboarding to the app easier for you?

#### **Overall**

- 1. How have you been using the app? How often?
- 2. Have you encountered any issues / problems with the app?

Study Protocol Form Version 7.4 Form Doc ID: AZDoc0059948 Parent Doc ID: SOP LDMS 001 00164328120

- a. How did you resolve the issue, if at all?
- 3. Overall, what do you think of the asthma app?
  - a. What parts are most / least useful?
- 4. Did it remind you of any other apps you've used before?

# **Specific Features**

[Explore use and satisfaction of the following app features]

Questions for below:

- -Did you use [feature]?
- -How useful/helpful or not is [feature]?
- -Any issues / problems with [feature]?
- -What could be done to make this [feature] better?

| Feature Set |
|--------------------------|
| Daily Log |
| Air Quality |
| Appointments |
| Asthma Control Test (ACT |
| Education |
| My Plan |
| Trends |
| Messaging |
| Notifications |

[Additional questions to probe on when exploring a given feature]

## 1. Daily log

- a. How often do you typically fill out your log?
  - i. What was your longest log streak?
- b. What time of day do you generally fill out the log? Why that time?
- c. Are there any questions in the daily log that are confusing? That do not apply to you?
  - i. Do you own a peak flow meter? Ability to record FEV1?
- d. Were the symptoms you were experiencing always reflected in the list of symptom options?
  - i. What about triggers?
- e. To what extent did the medication question make sense? Is 'Quick-relief / asneeded' a familiar term?
- f. How helpful was the review screen?
- g. How often did you go back and add a log for days that you missed?
- h. How often did you go back in and edit logs?
- i. How, if at all, do you know that a clinician is looking at your log data?
- j. Do you have any thoughts on how we can make filling out the log easier for you?

## 2. Air Quality

- a. How important is air quality to track for you?
- b. Is this something you tracked prior to the app?
- c. How else did you use this feature i.e., did you use it to track allergens like pollen, ragweed, etc.?
  - i. If yes, how helpful? If no, why not?

## 3. Appointments

- a. How accurate was the information reflected in the appointments card? Anything unusual?
- b. How many appointment reminders did you receive?
- c. Did you use the link to schedule additional appointments? Why/why not?

## 4. Asthma Control Test (ACT)

- a. How was this different from the daily log for you?
- b. How easy / difficult were the questions?
- c. Have you ever taken this questionnaire before?
- d. Why do you think your clinicians wanted you to answer these questions?

#### 5. Education

- a. Which articles did you explore if any?
  - i. Asthma EDU? Depression EDU?
- b. What education is missing that would be important to have?
- c. What type of media format do you prefer: video, articles, podcasts, etc.?

# 6. My Plan

- a. How helpful was it to have your list of medications available? How did you use it?
  - i. How accurate was the list of medications? How accurate were the images of your medications?
  - ii. Was there anything confusing about the list?
- b. Did you use the medication reminder feature? If so, how helpful was that?

## 7. Trends

- a. How did you use Trends?
  - i. To what extent did you use Trends in your appointment(s) with your doctor?
  - ii. Which view (daily, weekly) did you use the most?
- b. What do you think is the purpose of Trends?
- c. To what extent is this the type of information you are interested in seeing?
- d. How easy/difficult were the graphs to understand and interpret?
- e. Did you use the 'share with caregiver' feature? If so, who did you share with and why?

## 8. Messaging

- a. What types of messages did you send to your clinician?
  - i. Which subject line did you most commonly select?
- b. What was the response time like?
- c. How would you normally get in touch with your clinician before you had this app?

#### 9. Notifications

- a. What types of notifications did you receive from the app?
- b. How helpful were those notifications?
- c. Did you turn on/off any notifications? What did you think of the frequency?

## **Bugs / Reporting**

- 1. Have you encountered any bugs in the app?
  - a. [if yes] were you able to report the bug?
- 2. Did you have to contact the support team at all?
  - a. If so, how helpful were they?
  - b. Were they able to resolve the issue you had?

## **Appointments with Doctor**

- 1. Have you had any appointments with your doctor since you started using the app?
  - a. If yes, how if at all was that appointment different than what you're used to?
  - b. How if at all did they talk about the data that you put in the app?
  - c. At any point during the appointment, did you pull up your app to show them anything you had recorded?

#### Value

- 1. What have you gained, if anything, from using this app?
- 2. If you had a magic wand, what would you change about this app?
- 3. On a scale of 1 to 5 (1=not at all; 5=extremely), how likely would you be to recommend this app to someone else living with asthma?
  - a. Why a [#]?
  - b. [if less than 5] What would bring your score closer to a 5?

What else do you think the team should know about the app that we haven't already discussed here today?

# 25. APPENDIX P. RECRUITMENT TRACKING LOG

# RECRUITMENT TRACKING LOG (EVA-28838): SITE [XXX]

# Please send the Recruitment Tracking Log to Evidera via SharePoint

| Participant<br>ID | BI Linked ID | Patient<br>Age | Patient<br>Sex | Recruitment Quotas | Phone Type (Operation<br>System) | Outcome | Reason for Ineligible |
|---|---|---|---|---|---|---|---|
| | | | ⊠ Male □ Female | <ul> <li>New in practice (&lt; 3 months) but uncontrolled</li> <li>≥ one exacerbation in past 12 months</li> <li>Young adult</li> <li>Adult</li> </ul> | ☐ iOS (iOS 13 and iPhone 8 or newer) ☐ Android (OS 8.0 or newer) ☐ Other | ⊠ Eligible □ Ineligible □ Declined | |
| | | | ☐ Male ☐ Female | <ul> <li>New in practice (&lt; 3 months) but uncontrolled</li> <li>≥ one exacerbation in past 12 months</li> <li>Young adult</li> <li>Adult</li> </ul> | ☐ iOS (iOS 13 and iPhone 8 or newer) ☐ Android (OS 8.0 or newer) ☐ Other | ☐ Eligible ☐ Ineligible ☐ Declined | |
| | | | ☐ Male ☐ Female | <ul> <li>New in practice (&lt; 3 months) but uncontrolled</li> <li>≥ one exacerbation in past 12 months</li> <li>Young adult</li> <li>Adult</li> </ul> | ☐ iOS (iOS 13 and iPhone 8 or newer) ☐ Android (OS 8.0 or newer) ☐ Other | ☐ Eligible ☐ Ineligible ☐ Declined | |
| | | | ☐ Male ☐ Female | New in practice (< 3 months) but uncontrolled ≥ one exacerbation in past 12 months | ☐ iOS (iOS 13 and iPhone 8 or newer) ☐ Android (OS 8.0 or newer) ☐ Other | ☐ Eligible ☐ Ineligible ☐ Declined | |

Study Protocol Form Version 7.4

Form Doc ID: AZDoc0059948

Parent Doc ID: SOP LDMS\_001\_00164328124

| Study Protocol |
|------------------------------------|
| Study Code D2287R00166 [EVA-28838] |
| Version 7.4 |
| Date August 10, 2021 |

| ☐ Young adult |
|---------------|
| ☐ Adult |

Study Protocol Form Version 7.4

Form Doc ID: AZDoc0059948

Parent Doc ID: SOP LDMS\_001\_00164328125

## **26. SIGNATURES**

# **ASTRAZENECA SIGNATURE(S)**

# AMAZE Asthma Implementation clinical pilot Study - MGH

This Interventional Study Protocol has been subjected to an internal AstraZeneca review. I agree to the terms of this Study protocol.

AstraZeneca representative

<<*Name*, *title*>> Date

(Day Month Year)

<< Email address and telephone number>>

AstraZeneca representative

<<*Name*, *title*>> Date

(Day Month Year)

<< Email address and telephone number>>

This document contains confidential information, which should not be copied, referred to, released or published without written approval from AstraZeneca. Investigators are cautioned that the information in this protocol may be subject to change and revision.